Creation date: May 2018

Phase I clinical study, to evaluate the safety and tolerability of the preservative-free ophthalmic solution PRO-122 compared with Krytantek Ofteno®, elaborated by Sophia Laboratories, S.A. of C.V. on the ocular surface of ophthalmologically and clinically healthy subjects .

Protocol code: SOPH122-0518/I

Protocol version: 1

Date of the version: 22/05/2018

Registry: Pending

**Sponsor**: Sophia Laboratories, S.A. of C.V.



### 1. Summary.

#### 1.1 Synopsis.

#### Title of the study:

Phase I clinical study, to evaluate the safety and tolerability of the preservative-free ophthalmic solution PRO-122 versus Krytantek Ofteno®, elaborated by Sophia Laboratories, S.A. of C.V. on the ocular surface of ophthalmologically and clinically healthy subjects

| Protocol code: | Creation date: |
|---|---|
| SOPH122-0518/I | 22/05/2018 |
| Protocol version: | Date of the version: |
| 1 | 22/05/2018 |
| Therapeutic indication: | Use: |
| Ocular hypotensive | Primary open-angle glaucoma and ocular hypertension. |
| <b>Study period</b> (from the first visit of the first patient to the preparation of the final report): | Development phase: |
| 4 months | 1 |

#### **Objectives:**

To evaluate the safety and tolerability of the preservative-free formulation PRO-122 manufactured by Sophia Laboratories, S.A. of C.V. on the ocular surface of clinically healthy subjects.

#### **Hypothesis:**

The ophthalmic solution PRO-122 presents a profile of safety and tolerability similar to Krytantek Ofteno®, in healthy subjects.

#### Methodology:

Phase I clinical trial, controlled, parallel group, double blind, randomized.

| Number of patients: | Main inclusion criteria: |
|------------------------------------|------------------------------|
| n=24 | Clinically healthy subjects. |
| 12 subjects per group (both eyes). | |

#### Main selection criteria:

#### Inclusion criteria:

- Clinically healthy
- Ability to give your signed informed consent, and show willingness to comply with study procedures and to modify your lifestyle activities (Section 6.2.2)
- Age between 18 to 45 years.
- Indistinct sex.

- Women must ensure a hormonal contraceptive method or intrauterine device during the study period.
- Blood tests: within normal parameters or with a range of ± 20% as long as the subject is clinically healthy.
  - o Blood count (BH): Hemoglobin, erythrocytes, hematocrit, total leukocytes, platelets, mean corpuscular volume and mean corpuscular hemoglobin.
  - o Blood chemistry of three elements (QS): Glucose, urea and creatinine.
  - Liver function tests (PFH): TGO, TGP, total bilirubin, direct and indirect.
- Visual ability 20/30 or better in both eyes.
- Vital signs within normal parameters.
- Intraocular pressure ≥10 and ≤ 21 mmHg.

#### Exclusion criteria:

- Users of topical ophthalmic products of any kind.
- Users of medicines, or herbal products, by any other route of administration, with the exception of hormonal contraceptives in the case of women.
- Women who are pregnant or breastfeeding.
- Participation in clinical research studies 90 days prior to inclusion in the present study.
- Previous participation in this same study.
- Users of contact lenses.
- History of any chronic-degenerative disease.
- Inflammatory or infectious disease, active at the time of study entry.
- Injuries or traumatisms not resolved at the time of admission to the study.

#### Test product, dose and route of administration:

- PRO-122. Timolol 0.5% / brimonidine 0.2% / dorzolamide 2% ophthalmic solution free of preservatives. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
- Dosage: 1 drop every 12 hours, in both eyes
- Route of administration: topical ophthalmic.

#### Test product, dose and route of administration:

- 1. Krytantek Ofteno<sup>®</sup>. Timolol 0.5% / brimonidine 0.2% / dorzolamide 2% ophthalmic solution. Prepared by Sophia Laboratories, S.A. of C.V., Zapopan, Jalisco, Mexico.
- Dosage: 1 drop every 12 hours, both eyes.
- Route of administration: topical ophthalmic.

| Treatment duration: | Duration of subject in the study: |
|---------------------|-----------------------------------|
| 7 days. | 15 to 22 days. |

#### **Evaluation criteria:**

#### **Primary outcome variables:**

- o Incidence of adverse events (Time of Evaluation: day 4, 8 and 14).
- Ocular Comfort Index (ICO) score (TE: day 8).

#### Secondary outcome variables:

- Changes in visual ability (TE: day 4 and 8).
- Changes in corneal and conjunctival staining with lysine green (TE: day 4 and 8).
- Changes in corneal and conjunctival staining with fluorescein (TE: day 4 and 8).
- Conjunctival hyperemia changes (TE: day 4 and 8).

- o Incidence of chemosis (TE: day 4 and 8).
- o Incidence of alterations in the results of laboratory tests (TE: day 8).
- o Incidence of alterations in heart rate (TE: day 4 and 8).
- Incidence of alterations in the respiratory frequency (FR) (ET: day 4 and 8).
- o Incidence of alterations in systemic blood pressure (SBP) (TE: day 4 and 8).

#### **Exploratory outcome variables:**

Changes in intraocular pressure (ET: day 4 and 8).

#### Statistical methodology:

The data will be expressed with measures of central tendency: mean and standard deviation for the quantitative variables. The qualitative variables will be presented in frequencies and percentages. The statistical analysis will be carried out by means of the Mann-Whitney U test for the quantitative variables for the difference between the groups. The difference between the qualitative variables will be analyzed by means of X2 (Chi2). An alpha  $\leq$  0.05 will be considered significant.

## 1.2 Diagram of the study.



<sup>\*</sup> Baseline measurements can be taken from those made during the screening visit. It is the investigator's prerogative to perform them again at the baseline visit.

# 1.3 Schedule of the study.

| Procedures | Scrutiny | VB | V1 | VF | LIS |
|---|---|---|---|---|---|
| Procedures | D 1 - Xª | D 0 | D 4 ± 1 | D 8 to + 1 | D 14 ± 1 |
| CI Signature | Х | | | | |
| Clinic history | Χ | | | | |
| Blood sampling | Χ | | | Χ | |
| Urine pregnancy test | Χ | | | Χ | |
| PIO | Χ | X <sup>1</sup> | Х | Χ | |
| CV | Χ | X <sup>1</sup> | Х | Χ | |
| Ocular surface stains | Χ | X <sup>1</sup> | Х | Χ | |
| Comprehensive ophthalmological evaluation | X | X <sup>1,2</sup> | Х | X <sup>2</sup> | |
| Vital signs | Χ | X <sup>1</sup> | Χ | Χ | |
| Eligibility criteria | Χ | $X_p$ | | | |
| EA evaluation | Χ | Χ | Χ | Χ | Χ |
| Review of laboratory results | | Х | | | Χ |
| IP Assignment | | Xc | | | |
| MC evaluation | | Х | Х | Χ | |
| Delivery of the IP and start of intervention | | X | | | |
| Ocular Comfort Index | | Х | | Х | |
| Adherence evaluation | | | Χ | Χ | |
| Daily delivery of the subject | | Х | Х | | |
| Continuity evaluation of the subject | | | х | | |
| Return / Evaluation of the subject's Journal | | | х | Х | |
| Return of IP | | | | Χ | |

a The counting visit may be up to 7 days before the baseline, if it exceeds these the subject can not enter.

b These criteria will be completed with the results of the laboratory tests and those obtained during the screening visit.

C Indication to start application the next day

<sup>1</sup> They can be taken from the scrutiny visit, it is the prerogative of the PI to measure them again at the baseline visit.

<sup>2</sup> Includes subsequent segment valuation

# Page intentionally left blank

# 2. Content.

| <u>1.</u> | SUMMARY. | 1 |
|---|---|---|
| 1.1 | Synopsis. | 1 |
| 1.2 | DIAGRAM OF THE STUDY. | 4 |
| 1.3 | SCHEDULE OF THE STUDY. | 5 |
| <u>2.</u> | CONTENT. | 7 |
| <u>3.</u> | INDEX OF ABBREVIATIONS. | 11 |
| <u>4.</u> | ADMINISTRATIVE STRUCTURE OF THE STUDY. | 13 |
| <u>5.</u> | INTRODUCTION. | 15 |
| 5.1 | THEORETICAL FRAMEWORK. | 15 |
| 5.2 | BACKGROUND. | 16 |
| 5.3 | STATEMENT OF THE PROBLEM. | 20 |
| 5.4 | JUSTIFICATION. | 20 |
| 5.5 | OBJECTIVES AND HYPOTHESES. | 21 |
| | 1 GENERAL OBJECTIVE. | 21 |
| | 1.1 Specific objectives. | 21 |
| | 2 SECONDARY OBJECTIVES. | 21 |
| | 3 EXPLORATY OBJECTS. | 21 |
| | 4 Hypothesis. | 21 |
| 5.6 | | 21 |
| | 1 DISCUSSION OF THE STUDY DESIGN. | 21 |
| 5.6. | 2 JUSTIFICATION OF THE POSOLOGY. | 22 |
| <u>6.</u> | MATERIAL AND METHODS. PARTICIPANTS, INTERVENTIONS AND VARIABLES. | 23 |
| 6.1 | STUDY CENTER. | 23 |
| 6.1. | 1 Organization of the center. | 23 |
| 6.1. | 2 DOCUMENTATION TO BE DELIVERED TO THE SPONSOR. | 23 |
| 6.1. | | 24 |
| | STUDY POPULATION. | 24 |
| | 1 Selection Criteria. | 24 |
| 6.2. | | 24 |
| | 1.2 Exclusion criteria. | 24 |
| | 1.3 Disposal criteria. | 25 |
| 6.2. | | 25 |
| 6.2. | | 25 |
| 6.2. | 4 RECRUITMENT AND RETENTION STRATEGIES. | 26 |

| 6.2.5 | IDENTIFICATION OF THE SUBJECT. | 26 |
|---|---|---|
| 6.3 I | NTERVENTION. | 27 |
| 6.3.1 | MEDICATIONS ADMINISTERED. | 27 |
| 6.3.1.1 | Drug under study. | 27 |
| 6.3.1.2 | Reference treatment. | 27 |
| 6.3.2 | STRATEGIES TO IMPROVE ADHERENCE AND PROCEDURE TO MONITOR ADHERENCE. | 28 |
| 6.3.2.1 | Procedure to monitor adherence. | 28 |
| 6.3.3 | TREATMENTS AND CONCOMITANT MEDICATIONS ALLOWED AND PROHIBITED DURING THE STUDY. | 29 |
| 6.3.4 | TREATMENT MANAGEMENT. | 29 |
| 6.3.4.1 | Delivery and reception. | 29 |
| 6.3.4.2 | Storage . | 30 |
| 6.3.4.3 | B Return. | 30 |
| 6.4 E | DELAY VARIABLES. | 30 |
| 6.4.1 | SECURITY VARIABLES. | 30 |
| 6.4.1.1 | Primary outcome variables. | 30 |
| 6.4.1.2 | 2 Variables of primary outcome of tolerability. | 30 |
| 6.4.1.3 | 3 Variables of secundary outcome | 30 |
| 6.4.2 | EXPLORATORY VARIABLES. | 30 |
| 6.4.3 | METHODS AND SCALES TO BE USED FOR THE MEASUREMENT OF THE VARIABLES. | 31 |
| 6.4.3.1 | Visual capacity. | 33 |
| 6.4.3.2 | 2 Comprehensive ophthalmologic evaluation. | 33 |
| 6.4.3.3 | B Eye comfort index. | 33 |
| 6.4.3.4 | Integrity of ocular surface: | 34 |
| 6.4.3.5 | Presence of adverse events. | 34 |
| 6.4.3.6 | 5 Intraocular pressure. | 34 |
| 6.4.3.7 | Vital signs. | 34 |
| 6.4.3.8 | B Laboratory tests. | 35 |
| 6.4.4 | MEASUREMENT TIME. | 35 |
| 6.5 T | IMELINE AND STUDY DIAGRAM. | 36 |
| 6.5.1 | PROCEDURES TO BE CARRIED OUT PER VISIT. | 37 |
| 6.5.1.1 | Scrutiny visit. | 37 |
| 6.5.1.2 | Baseline visit. | 37 |
| 6.5.1.3 | 3 Visit 1 | 38 |
| 6.5.1.4 | Final visit | 38 |
| 6.5.1.5 | Return of the IP: refers to the return by the subject, of the surplus IP, to the center. | 38 |
| 6.5.1.6 | Return / evaluation of the subject's diary: see Visit 1. | 38 |
| 6.5.1.7 | Adherence evaluation: refers to the assessment made by the PI according to section | |
| 6.3.2.1 | Procedure to monitor adherence. | 38 |
| 6.5.1.8 | Adverse events: see 6.4.3.5 Presence of adverse events. | 38 |
| 6.5.1.9 | Urine pregnancy test: see Screening visit. | 38 |
| 6.5.1.1 | .0 Vital signs: see 6.4.3.7 Vital signs. | 38 |
| 6.5.1.1 | .1 Visual capacity: see 6.4.3.1 Visual capacity. | 38 |
| 6.5.1.1 | .2 Comprehensive ophthalmological evaluation: see 6.4.3.2. Comprehensive | |
| ophtha | almological evaluation | 38 |
| 6.5.1.1 | .3 Integrity of the ocular surface: see 6.4.3.4 Integrity of ocular surface: | 38 |
| 6.5.1.1 | .4 Intraocular pressure: see 6.4.3.6 Intraocular pressure. | 38 |
| 6.5.1.1 | .5 Sampling of laboratory samples: see 6.4.3.8 Laboratory tests. | 38 |
| 6.5.1.1 | .6 Eye comfort index: see 6.4.3.3 Eye comfort index | 38 |

| 6.5.1.18 Security call. | 39 |
|--------------------------------------------------------------------|----|
| 6.5.1.19 Early termination visit. | 39 |
| 6.5.2 STUDY DIAGRAM. | 39 |
| 6.6 SAMPLE SIZE. | 40 |
| 6.6.1 CALCULATION OF THE SAMPLE SIZE. | 40 |
| 6.7 RECRUITMENT. | 41 |
| 7 METHODS ASSIGNMENT OF THE INTERVENTION | 42 |
| 7. METHODS. ASSIGNMENT OF THE INTERVENTION | 42 |
| 7.1 GENERATION OF THE ALLOCATION SEQUENCE. | 42 |
| 7.1 GENERATION OF THE ALLOCATION SEQUENCE. 7.2 BLINDING MECHANISM. | 42 |
| 7.3 IMPLEMENTATION | 42 |
| 7.4 BLINDING (MASKING). | 42 |
| 7.4.1 OPENING OF BLINDING. | 42 |
| 7.4.1 OPENING OF BLINDING. | 42 |
| 8. METHODS. COLLECTION, ADMINISTRATION AND DATA ANALYSIS. | 43 |
| 8.1 METHODS OF DATA COLLECTION. | 43 |
| 8.1.1 STRATEGIES TO COMPLETE THE FOLLOW-UP. | 43 |
| 8.2 DATA MANAGEMENT. | 43 |
| 8.3 STATISTICAL METHODOLOGY. | 44 |
| 8.3.1 Analysis of Primary and Secondary Outcome Variables. | 44 |
| 8.3.2 Additional analyzes. | 47 |
| 8.3.3 POPULATION ANALYSIS AND MANAGEMENT OF MISSING DATA. | 47 |
| 9. METHODS. MONITORING. | 48 |
| 9.1 DATA MONITORING. | 48 |
| 9.2 Adverse events. | 48 |
| 9.2.1.1 Record of adverse events in the Case Report Form. | 49 |
| 9.2.1.2 Follow-up of adverse events. | 50 |
| 9.2.1.3 Procedures for a serious adverse event. | 50 |
| 9.2.1.4 Causality assessment. | 52 |
| 9.2.2 RESPONSIBILITIES OF THE SPONSOR. | 53 |
| 9.3 UNANTICIPATED PROBLEMS. | 53 |
| 9.3.1 REPORT OF PNAS. | 53 |
| 9.4 Audit. | 54 |
| 9.4.1 Pre-study audit. | 54 |
| 9.4.2 AUDIT / INSPECTION DURING THE CONDUCTION OF THE STUDY. | 54 |
| 10. ETHICAL CONSIDERATIONS. | 55 |
| 10.1 Approved of Tue consumers | |
| 10.1 APPROVAL OF THE COMMITTEES. | 55 |
| 10.2 AMENDMENTS TO THE PROTOCOL. | 55 |
| 10.3 EARLY TERMINATION OF THE STUDY. | 56 |

| 10.4 CONSENT. | 57 |
|-----------------------------------------------------|----|
| 10.4.1 Obtaining. | 57 |
| 10.4.2 Special considerations. | 57 |
| 10.4.3 MODIFICATION TO INFORMED CONSENT. | 57 |
| 10.5 CONFIDENTIALITY. | 58 |
| 10.6 CONFLICT OF INTERESTS. | 58 |
| 10.6.1 Declaration of interests. | 58 |
| 10.7 Access to information. | 59 |
| 10.8 AUXILIARY CARE AND AFTER THE END OF THE STUDY. | 59 |
| 10.9 BIOSECURITY ASPECTS. | 59 |
| 10.10 FINAL REPORT AND PUBLICATION OF RESULTS. | 59 |
| 10.10.1 Final report. | 59 |
| 10.10.2 COMMUNICATION OF RESULTS. | 59 |
| 10.10.3 PUBLICATION OF RESULTS. | 59 |
| 11. BIBLIOGRAPHIC REFERENCES. | 61 |
| 12. SIGNATURE PAGE. | 65 |
| 12.1 SIGNATURES OF THE SPONSOR'S REPRESENTATIVES. | 65 |
| 12.2 Investigator. | 65 |
| 13. ANNEXES. | 67 |
| 13.1 OCULAR COMFORT INDEX. | 67 |
| 13.2 EFRON SCALE FOR CONJUNCTIVAL HYPEREMIA. | 68 |
| 13.3 Oxford Scale. | 68 |

# 3. Index of abbreviations.

AA alpha-adrenergic agonist

**ALT** Alanine transferase

AST Aspartate transferase

BAK Benzalkonium chloride, (for its acronym in English Benzalkonium chloride.)

BB Betablocker

BD Bilirubin direct

BI Bilirubin indirect

BH Blood count

**BPC** Good clinical practices

BT Total Bilirubin

CV Visual capacity

IEC Research Ethics Committee

CI Informed Consent

CCI informed consent letter

CRF Case Report Form (Case Report Form)

EA / EAS Adverse event / serious adverse event

FDA Food and Drug Administration (Food and Drug Administration)

FC Heart rate

FR Respiratory frequency

GPAA Primary open angle glaucoma

HTO Intraocular hypertension

IAC Carbonic anhydrase inhibitors

PRO-122

ICH International Harmonization Conference (International Conference on

Harmonization)

ICO Eye comfort index

IP study medication

IOP intraocular pressure
PFH Liver function tests

PGA Prostaglandins Analog

PI Principal investigator of the clinical study

QS Blood chemistry

TAS Systemic blood pressure

TE Scan time

TF Fluorescein staining

TMMT Maximum tolerated medical therapy

TVL Green lysine stain

### 4. Administrative structure of the study.

The administrative structure of the sponsoring party, corresponding to Sophia Laboratories, S.A. of C.V. is shown in **Table 1. Administrative structure** 

| Function | Name/Contact | Affiliation ¥ |
|---|---|---|
| Medical responsible for the study | Dr. Leopoldo Martín Baiza Durán leopoldo.baiza@sophia.com.mx | Medical Director and Regulatory<br>Affairs |
| Director of the study | QFB. Francisco García Vélez francisco.garcia@sophia.com.mx | Clinical Operations Manager |
| Clinical Team | Dr. Oscar Olvera Montaño oscar.olvera@sophia.com.mx | Medical Editor |
| Clinical Team | Dr. in C. Ricardo Alonso Llamas Velázquez ricardo.llamas@sophia.com.mx | Clinical Security Pharmacologist |
| Clinical Team | Dra. in C. Patricia del Carmen Muñoz Villegas patricia.munoz@sophia.com.mx | Biostatist |

Employees of Sophia Laboratories, S.A. of C.V Av. Paseo del Norte No.5255, Col. Guadalajara Technology Park, Carretera Guadalajara-Nogales Km13.5 C.P. 45010 Zapopan, Jalisco, Mexico Tel +52 (33) 3000 4200.

Table 1. Administrative structure.



Figure 1. Administrative structure of the study.

# Page intentionally left blank

#### 5. Introduction.

#### 5.1 Theoretical framework.

Glaucoma is a progressive optic neuropathy characterized by the loss of ganglion cells of the retina and their respective axons, resulting in the distinctive appearance of the optic disc and concomitant loss of visual function. [1] It is the second cause of blindness worldwide and it is estimated that by 2020, 79.6 million people will have glaucoma, with 74% of these corresponding to primary openangle glaucoma (POAG). [2] The Latin American population, especially that of Mexican origin, is more prone to develop POAG compared with whites. [3, 4]

The mechanism by which glaucoma damages the optic nerve is probably multifactorial, notwithstanding, elevated intraocular pressure (IOP) is the main risk factor and the only one that can be modified at present to prevent the progression of glaucoma damage, including Normo-tense glaucoma. [5, 6, 7, 8, 9]. It has also been shown that the reduction in IOP decreases the rate of conversion of ocular hypertension (OHT) to glaucoma. [7] Chauhan et al have reported that for every 1 mmHg increase in IOP, the risk of glaucoma progression increases 19%. [5]

Despite the great advances in surgical filtering treatments, implants and laser procedures that improve trabecular drainage, pharmacological therapy continues to be the initial intervention for the majority of patients with OHT and glaucoma; this treatment typically includes the topical application of antihypertensive agents. [10]

Currently the pharmacological options for the reduction of IOP, with topical application, include prostaglandin analogues (PGA), beta blockers (BB), alpha adrenergic agonists (AA), carbonic anhydrase inhibitors (CAI) and parasympathomimetics. Commonly, pharmacotherapy begins with the application of a single hypotensive agent, usually of the so-called first line (prostaglandin analogs or beta blockers). [11] Nevertheless, monotherapy may be insufficient in many cases, due to the inability to reach the target IOP and / or prevent the progression of glaucoma. In some other cases, the same medication may lose its effectiveness over time, due to tachyphylaxis. [12] The Ocular Hypertensive Treatment Study reported that at 5 years, about 40% of patients require two medications to achieve a 20% reduction in IOP compared to baseline, while an additional 9% needs more than two medications. [7] Therefore, more than one medication is frequently required for the adequate control of IOP in the medium and long term. This can be achieved with the concurrent use of two or more drugs of different classes, either by its concomitant application or in a fixed combination. [12]

In addition to the effectiveness in decreasing IOP, fixed combinations offer multiple benefits when compared with the concomitant application of their active principles. [13] These benefits include lower cost, simpler treatment regimen, better adherence to treatment and decreased risk of washing. [14, 15]

Fixed combinations also offer a decrease in the risk of corneal damage and ocular surface associated with cumulative exposure of preservatives. For example, chronic exposure to benzalkonium chloride (BAK), used in many ophthalmological drugs, has been associated with inflammation and conjunctival and corneal damage, alterations of the tear film and symptoms of ocular surface disease. [16, 17, 18]

Currently the fixed combinations available include BB timolol 0.5% combined with a drug from the other therapeutic families, a PGA, an AA or a topical ICA. [19] In Mexico and other South American

Version 1

countries there is also the triple fixed combination, which includes timolol, brimonidine and dorzolamide.

#### 5.2 Background.

The preservatives are used with the purpose of inhibiting the microbial growth and suppressing biodegradation inside the medicines. [20] A variety of conservatives have been used throughout history. The chronic use of these drugs has been linked to irritation and alterations of the ocular surface, it has been established that the conservatives themselves have adverse events, which are attached to those of the active principle that preserve. [21]

The preservatives are classified into detergents and oxidants, and a more recent version of oxidants called buffered by ions. [20] BAK is the most historically used preservative, belongs to the class of detergents and its concentration in ocular hypotensives varies from 0.004 to 0.02%, the reasons for its popularity include its broad spectrum of action and its familiarity with the formulating industry. While its effectiveness is well recognized, there are numerous studies documenting the harmful effects of BAK. It is known that BAK at concentrations of 0.05-0.1% induces necrosis and at concentrations of 0.01% apoptosis. Its effects are cumulative and become more severe at higher concentration and with more frequent exposures. [20, 22]

The triple fixed combination has been evaluated in several studies, being compared against double fixed combinations. In a randomized, double-blind study in 112 patients, the IDB application was compared for 180 days of fixed triple therapy against the 0.5% timolol / fixed 2% dorzolamide combination. The triple combination was superior with a difference of 3.4mmHg in the average IOP in the third month. [23]

Another study compared the tripla fixed combination against the fixed combination timolol 0.5% / brimonidine 0.2%. It was a double blind, randomized study in patients with glaucoma and / or ocular hypertension, with BID application for 3 months. The triple combination was superior with a difference of 2.16mmHg in the average IOP at the third month in the 08:00 hours review. [24]

*Baiza L et al.*, Conducted a study in which evaluated the safety profile of the ophthalmic solution consisting of 0.5% timolol / 2% dorzolamide / brimonidine versus the ophthalmic solution constituted by timolol / dorzolamide in patients with primary open angle glaucoma and / or intraocular hypertension who received for 6 months 1 drop BID of the product under investigation and comparator drug.

Results: 112 patients participated in the study, who were divided into 2 study groups, 56 subjects for each pharmacological intervention. Regarding the safety profile: there were no significant differences in the parameters of visual acuity, hyperemia, stains, visual fields, symptomatology (eye pain, burning, photophobia and foreign body sensation) between the study groups. Group exposed to timolol / dorzolamide / brimonidine: 2/56 (3.5%) subjects reported presenting at least 1 adverse event. In the group that received timolol / dorzolamide, 6/56 subjects were registered who manifested at least 1 adverse event. None of the events that occurred motivated the removal or elimination of any patient. The research group concluded that both the investigational product and the comparator drug were safe and well tolerated. It showed better safety profile with the triple combination. (Table 3. Adverse events of the Baiza study 2009) [25]

| Adverse event | Brimonidine / brinzolamide<br>N= 435<br>n (%) | Brinzolamide<br>N= 460<br>n (%) | Brimonidine<br>N= 455<br>n (%) |
|---|---|---|---|
| Ocular | | | |
| Blurry vision | 23 (5.3%) | 30 (6.5%) | 1 (0.2%) |
| Eye irritation | 18 (4.1%) | 6 (1.3%) | 10 (2.2%) |
| Eye allergy | 11 (2.5%) | 0 (0%) | 5 (1.1%) |
| Ocular hyperemia | 9 (2.1%) | 3 (0.7%) | 15 (3.3%) |
| Eye pain | 9 (2.1%) | 8 (1.7%) | 5 (1.1%) |
| Allergic conjunctivitis | 8 (1.8%) | 2 (0.4%) | 7 (1.5%) |
| Eye itching | 7 (1.6%) | 5 (1.1%) | 3 (0.7%) |
| Conjunctival hyperemia | 7 (1.6%) | 5 (1.1%) | 5 (1.1%) |
| Dry Eye | 6 (1.4%) | 4 (0.9%) | 7 (1.5%) |
| Conjunctivitis | 6 (1.4%) | 1 (0.2%) | 8 (1.8%) |
| Foreign body sensation | 5 (1.1%) | 3 (0.7%) | 2 (0.4%) |
| No ocular | | | |
| Dysgeusia | 17 (3.9%) | 38 (8.3%) | 1 (0.2%) |
| Dry mouth | 13 (3.0%) | 0 (0%) | 11 (2.4%) |
| Fatigue | 3 (0.7%) | 0 (0%) | 6 (1.3%) |

Table 2. Adverse events in the Realini study.

| Adverse event | Timolol / brimonidine /<br>dorzolamide group<br>N=56 | Group<br>timolol / dorzolamide<br>N=56 |
|---|---|---|
| Eye pain | 1 | - |
| Burning and eye pain | 1 | - |
| Eye pain and headache | - | 1 |
| Keratitis and eye pain | - | 2 |
| Keratitis and chemosis | - | 1 |
| Keratitis and burning | - | 1 |
| Burning | - | 1 |

Subjects who manifested at least 1 adverse event during their participation in the study.

Table 3. Adverse events of the Baiza study 2009.

In another study conducted by the research team of Baiza L, et al, the safety profile of the combined fixed therapy was determined in ophthalmic solution, constituted by 0.5% timolol / 0.2% brimonidine / dorzolamide 2% versus one made up of timolol 0.5% / brimonidine 0.2% in patients with primary open-angle glaucoma and / or ocular hypertension who were divided into 0.5%

groups, which received 1 drop of the drug product or product in IDB research for 3 months. Results: 112 subjects participated, 56 patients per group. During the development of the study, no participant presented any serious adverse event. Of the total number of participants, only 8 reported having presented at least 1 non-serious adverse event. 6 subjects were withdrawn from the study, due to the development of adverse events. 2 people with ocular burning, one of mild intensity and one of moderate intensity, severe itching in one subject, foreign body sensation of mild intensity in one participant, red eye of severe intensity in another patient, severe dizziness in another patient, mild headache in another participant and mild intensity bradycardia in one more.

| Adverse event | Timolol / brimonidine /<br>dorzolamide group<br>N=56 | Group<br>timolol / brimonidine<br>N=56 |
|---|---|---|
| Ocular burning | 1 | 1 |
| Itch | 1 | - |
| Foreign body sensation | 1 | - |
| Red eye | - | 1 |
| Dizziness | - | 1 |
| Headache | - | 1 |
| Bradycardia | - | 1 |

Subjects who presented at least 1 adverse event during their participation in the study.

Table 4. Adverse events of the Baiza study 2012.

The research team concluded that the safety profile of the ophthalmic solution consisting of brimonidine, timolol and dorzolamide was better, because there were only 3 events compared to the 5 registered in patients who received dual therapy. Notwithstanding, both therapies were considered safe. [24] (Table 4. Adverse events of the Baiza study 2012)

García A, et al., Reported the safety profile by developing a cross-over clinical trial, 2 periods, 2 sequences involving patients with primary open-angle glaucoma and / or ocular hypertension who previously received the ophthalmic solution in combination fixed, conformed by bimatoprost 0.03% / timolol 0.5% or the ophthalmic solution in fixed combination constituted by brimonidine 0.2% / timolol 0.5% / dorzolamide 2% at a dose of 1 drop 2 times a day for 3 months; in each period, in the case of subjects exposed to triple therapy and a dose of 1 drop 1 time a day for 3 months; in each period, in the case of patients with combined double therapy.

Results: Few adverse events were reported by the participants throughout the study. The most frequent event was hyperemia and was the only event associated with the investigational drug. [27]

| Adverse event | Timolol / brimonidine /<br>dorzolamide group<br>N=78 | | Group<br>timolol / bimatoprost<br>N=78 |
|---|---|---|---|
| Vitreous hemorrhage | | 1 | |
| Pruritus | | 1 | |
| Severe hyperemia * | 1 | | 2 |
| Foreign body sensation and conjunctival edema * | - | | 1 |
| Severe eyelid edema | | 1 | |
| Reduction of the visual field * | 1 | | - |
| Allergy | | 1 | |
| Visual acuity decreased significantly | | 1 | |
| Blurry vision | | 1 | |
| Not specified* | 1 | | - |

Events reported in patients during the 6-month study. In total, 12 patients presented at least 1 adverse event, of which 6 subjects had to be removed from the research protocol due to the severity and seriousness of the event. \* Subjects removed from the study.

Table 5. Adverse events of García's study.

As can be seen in **Table 5. Adverse events of García's study** shows the event that occurred in the totality of the population evaluated during the development of the study, nevertheless, it refers to the type of intervention that the participant received at the time of presentation of the event that led to the patient's withdrawal.

Adverse reactions associated with 0.5% timolol maleate at ocular level may be: transient burning, decreased corneal sensitivity, allergic blepharoconjunctivitis, superficial punctate keratitis, conjunctival hyperemia, keratoconjunctivitis sicca, ptosis, diplopia, blurred vision, refractive changes (due, in some cases, to the suspension of treatment with miotics). At the level of the central nervous system: headache, dizziness, lethargy, confusion, hallucinations, fatigue and depression. Cardiovascular: systemic arterial hypotension, bradycardia, arrhythmia, atrioventricular heart block, cardiac arrest, congestive heart failure, syncope, stroke, tachycardia and cerebral ischemia; the latter have been more common in the elderly or in people with previous cardiovascular disorders. Adverse reactions at the respiratory level: bronchial spasm, (especially in subjects with a history of bronchospastic disorders), respiratory insufficiency and dyspnea. Other reactions: worsening of myasthenia gravis, alopecia, ungueal pigmentary changes, nausea, localized and generalized skin rash, urticaria, asthenia, sexual dysfunction, including impotence, decreased libido and reduced ejaculation; hyperkalemia, masking of symptoms of hypoglycemia in patients with insulindependent diabetes, diarrhea and paresthesias. [28]

The adverse reactions reported with the use of brimonidine tartrate 0.2%, in greater frequency are: dry mouth sensation, drowsiness, fatigue, cardiopulmonary alterations. At the ocular level: hyperemia, burning, blepharoconjunctivitis and allergic conjunctivitis, acute ocular conjunctivitis, transient miosis in people sensitive to the formula. [29]

Version '

Dorzolamide hydrochloride 2% is generally well tolerated. The most frequently reported adverse effects have been transient ocular burning, taste distortion, corneal erosion, conjunctival injection, blurred vision, lachrymation and ocular itching. [30]

#### 5.3 Statement of the problem.

For the treatment of HTO and GPAA, the use of a single medication may be insufficient when trying to reach the goal IOP, so it is necessary to resort to the use of 2 or more ocular hypotensives from different families. In a simplified scheme of treatment of glaucoma, it is proposed to start with monotherapy, based on a first line medication such as a PGA or a BB, the first being the most favored by ophthalmologists at present. If this initial therapy is not enough, but if it responds, a second medication is added, preferably the other first-line medication not previously used. In this intermediate therapy, the patient would already be receiving 3 to 4 daily instillations, theoretically compromising their attachment to the treatment and exposing it to a higher cumulative dose of BAK. So the attending physician may decide to migrate to a fixed combination of two medications. If the IOP goal is not achieved, a third medication can be added by reaching the maximum tolerated medical therapy scheme (TMMT) stipulated by Zimmerman of 3 medications in 3 daily instillations. [31]

As previously stated, the use of fixed combinations has advantages over the concomitant application of its components. As far as we know, there are no reports of the evaluation of the triple fixed combination compared to the concomitant application of its components. Fixed triple therapy can increase adherence to treatment with TMMT and broadens the horizon towards the new TMMT plan postulated by Sampaolesi, which includes fixed triple therapy + a PGA. [31]

#### 5.4 Justification.

During the treatment of a patient with glaucoma, it may be necessary, at some point in the evolution, to require 2 or more medications to achieve the desired control of IOP. Fixed combinations offer multiple advantages, including a simplified regimen that can lead to better attachment, greater convenience for the patient resulting from the use of fewer bottles and instillations, less exposure to preservatives that can potentially damage the ocular surface, eliminates the washing effect and finally an economical saving in the cost of the therapy.

In Mexico, since 2007, and in more recent years in other Latin American countries such as Bolivia, Colombia, Costa Rica, Ecuador, El Salvador, Guatemala, Honduras, Panama, Peru, the Dominican Republic and Uruguay, Krytantek Ofteno® is commercially available. Sophia Laboratories, S.A. of C.V., which is the fixed combination of Timolol 0.5% / Brimonidine 0.2% / Dorzolamide 2% in ophthalmic solution. During these years, Krytantek Ofteno® has shown its efficacy in the clinical practice of ophthalmologists who use it and its safety profile has been known through pharmacovigilance systems.

PRO-122 is a free reformulation of conservators of Krytantek Ofteno®, from which it is required to document its safety profile.

PRO-122

Version 1

#### 5.5 Objectives and hypotheses.

#### 5.5.1 General Objective.

To evaluate the safety and tolerability of the preservative-free ophthalmic solution PRO-122 on the ocular surface.

#### 5.5.1.1 Specific objectives.

- To compare the safety of the ophthalmic solution PRO-122 with Krytantek Ofteno® by means of the incidence of adverse events during the study.
- To compare the tolerability of the ophthalmic solution PRO-122 with Krytantek Ofteno® by means of the ICO score.

#### 5.5.2 Secondary objectives.

- Compare the safety of PRO-122 with Krytantek Ofteno® through changes in visual ability during visits.
- To compare the safety of PRO-122 with Krytantek Ofteno® through changes in corneal and conjunctival stains with lysine green during visits.
- To compare the safety of PRO-122 with Krytantek Ofteno® through changes in corneal and conjunctival stains with fluorescein during visits.
- To compare the safety of PRO-122 with Krytantek Ofteno® through changes in conjunctival hyperemia during visits.
- Compare the safety of PRO-122 with Krytantek Ofteno® by the incidence of chemosis during visits.
- To compare the safety of PRO-122 with Krytantek Ofteno® by means of the incidence of alterations in the results of the laboratory tests on day 11.
- To compare the safety of PRO-122 with Krytantek Ofteno® by the incidence of alterations in HR during visits.
- To compare the safety of PRO-122 with Krytantek Ofteno® by means of the incidence of alterations in RF during visits.
- To compare the safety of PRO-122 with Krytantek Ofteno® by the incidence of changes in SAD during visits.

#### 5.5.3 Exploraty objects.

Compare the changes in intraocular pressure during the visits.

#### 5.5.4 Hypothesis.

HO The ophthalmic solution PRO-122 presents a safety and tolerability profile similar to Krytantek Ofteno® in healthy subjects

Ha The ophthalmic solution PRO-122 presents a different safety and tolerability profile Krytantek Ofteno® in healthy subjects.

#### 5.6 Design and plan of the study.

Clinical trial, phase I, controlled, parallel group, double blind randomization, exploratory.

#### 5.6.1 Discussion of the study design.

The design of the study (clinical trial) is considered the highest standard of data quality when looking to explore the effect of an intervention. The phase of pharmacological development (phase I) corresponds to the objective of the study which is to assess the safety and tolerability, so that the intervention time is short and the sample size required is less than that of an efficacy clinical trial. The presence of parallel groups allows the comparison between the intervention groups on the

Version 1

outcome variables. Blinding and randomisation allow to reduce biases that are incurred with other designs, eg. Selection bias, evaluation bias, among others.

The comparator, Krytantek Ofteno®, has a known safety profile and shares the same active principles in the same concentrations as PRO-122, reason why it was chosen as an option to compare.

#### 5.6.2 Justification of the posology.

The chosen dosage is one drop every 12 hours, this is the approved dosage for the reference medicine. For this phase I study, we do not consider it necessary to expose the research subjects to dosage rates higher than those recommended, since it is not justifiable.

Version 1

# 6. Material and methods. Participants, interventions and variables.

#### 6.1 Study center.

The present study will be carried out in a research center previously evaluated by the sponsor. This center will be an institution or establishment where health research is carried out that complies with current regulations.

#### 6.1.1 Organization of the center.

Each study center will have a principal investigator (PI). The PI is the ophthalmology specialist responsible for the clinical study.

The PI will also be responsible for forming a multidisciplinary research team to carry out the clinical study according to protocol, under its scientific guidance. It is the prerogative of the PI the design of the organization of its center and the selection of the personnel that will perform the functions. However, the minimum organization of the research team requested by the sponsor requires the figure of sub-researcher, study coordinator and pharmacist or unblinded staff (See Figure 2 Minimum organization of the center).

Any person to whom the PI designates, under his / her responsibility, a part of the follow-up of the study (co-investigator, sub-researcher, nurse, etc.) or a specific function of participation in the study (pharmacist, administrative assistant, study coordinator, etc.) must appear in the "Delegation of Responsibilities" format.



Figure 2 Minimum organization of the center.

The "Delegation of Responsibilities" and the "Organizational Chart of the Center" must be delivered to the sponsor before the start of the study and updated if the members or their responsibilities are changed.

#### 6.1.2 Documentation to be delivered to the sponsor.

The PI must deliver to the sponsor, before the start of the study:

- Curriculum vitae updated, in Spanish, dated and signed (maximum 10 pages), of the PI and the personnel that make up the organizational chart of the center.
- Copy of PI academic certifications (degree certificate and specialty diploma in ophthalmology; federal professional certificates)
- Copy of academic certifications of the maximum degree obtained, from each one of the members of your research team, which cover their capacity to perform the delegated functions.

Clinical Trial Protocol: SOPH122-0518 / I

PRO-122

Version 1

- Copy of operation notice or similar issued by corresponding regulatory entity (When applicable)

Certificate of Good Clinical Practices in force. In case the certificate does not specify the validity time in the certificate, the date of issue of the certificate must not exceed one year.

#### 6.1.3 Closure of the center.

The closing of the center will be carried out once the last visit of the last included subject previously agreed between the sponsor and the PI has been made. The closing process will be according to the normal procedures of the sponsor's internal operations and must have the disposition and participation of the PI and whoever he designates.

It is the sponsor's prerogative to prematurely close a study center, it must inform the PI the reasons for the closure. These can be, but do not exclude:

- a) Less recruitment to the projected.
- b) Deviations greater than the protocol, which at the sponsor's discretion merit closing the center.
- c) Recidivism of deviations to the protocol, which at the sponsor's discretion merit closing the center.
- d) Early termination of the study.

#### 6.2 Study population.

#### 6.2.1 Selection criteria.

#### 6.2.1.1 Inclusion criteria.

- Be clinically healthy.
- Ability to grant signed informed consent and show willingness to comply with study procedures
- Have an age between 18 to 45 years.
- Indistinct sex
- Women must ensure a hormonal contraceptive method or intrauterine device during the study period.
- Presenting blood tests: within normal parameters or with a range of ± 20% as long as the subject is clinically healthy.
  - o Blood count (BH): Hemoglobin, erythrocytes, hematocrit, total leukocytes, platelets, mean corpuscular volume and mean corpuscular hemoglobin.
  - o Blood chemistry of three elements (QS): Glucose, urea and creatinine.
  - Liver function tests (PFH): TGO, TGP, total bilirubin, direct and indirect.
- Present visual ability 20/30 or better in both eyes.
- Present vital signs within normal parameters.
- Present intraocular pressure ≥10 and ≤ 21 mmHg.

#### 6.2.1.2 Exclusion criteria.

#### 6.2.1.2.1 General criteria.

Be a user of ophtalmic topical products of any kind.

- Be a user of medicines, or herbal products, by any other route of administration, with the exception of hormonal contraceptives in the case of women.
- In case of being a woman, being pregnant or breastfeeding.
- To have participated in clinical research studies 90 days prior to inclusion in the present study.
- Have previously participated in this same study.
- Be a user of contact lenses and can not suspend their use during the study.
- That they can not follow the lifestyle considerations described in the numeral 6.2.2

#### 6.2.1.2.2 Medical and therapeutic criteria.

- Having a history of any chronic degenerative disease.
- Presenting inflammatory or infectious disease, active at the time of study entry.
- Presenting unresolved injuries or traumas at the time of entering the study.

#### 6.2.1.3 Disposal criteria.

- Withdrawal of the consent letter under information.
- Presentation of a serious adverse event related or not to the investigational product, which
  has criteria of the PI and / or the sponsor could affect the ability of the patient to continue
  with the study procedures safely.
- No tolerability or hypersensitivity to any of the compounds used during the tests (fluorescein, green lysine, tetracaine)
- No tolerability or hypersensitivity to any of the investigational drugs.

#### 6.2.2 Lifestyle considerations.

For the study it is necessary that the participants modify the following activities of their lifestyle:

- Refrain from alcohol consumption, from entering the study to taking laboratory tests of the final visit.
- Refrain from tobacco use.
- Refrain from the use of electronic vaporizers.
- Avoid submerging in water without eye protection (goggles-protective glasses).
- Avoid direct exposure to fans (including air conditioning vents) during activities that involve sight. 24 hours before your review visits.
- Do not modify your sleep-wake cycle with which you enter the study.

#### 6.2.3 Scrutiny failures.

A failure to scrutinize is defined as those participants who agree to participate in the study, granting their consent, but who are not assigned to any intervention, that is, they do not enter the study. It is necessary that the following information of the inclusion faults be reported minimally:

- Demographic data
- Details of the scrutiny failure (specify if it is due to the eligibility criteria, to which, or some other reason for the failure).
- Presence of serious adverse events during the scrutiny.

The above is necessary to comply with the CONSORT (Consolidated Standards of Reporting Trials) guidelines for the publication of results or to answer possible questions from the regulatory authorities.

Subjects who do not meet the eligibility criteria to participate in the study (inclusion failure) due to a specific modifiable factor, could re-participate in the scrutiny. The subjects in this case must use the same initial counting number.

#### 6.2.4 Recruitment and retention strategies.

This is a phase I study, which will be conducted in a center. The selected center will be responsible for the recruitment of healthy subjects. The minimum recruitment index is 0.53 patients per day, because it must recruit 24 subjects in 45 days.

The duration of the participation of the subject in the study is short, so no retention problems are anticipated. However, the subjects will be creditors of a travel allowance support and fulfill their visits. Other strategies to improve the retention of subjects include, but are not limited to:

- Clearly inform the importance of the study and the benefits that the population will obtain from the results of the study.
- Make calls or send text messages to remember appointments or activities to perform.
- Provide a printed calendar and an identification card in order to remember appointments and activities that will be carried out, in addition to the estimated duration of the same.
- In case the participant does not attend his / her appointment, the research center must make a call to know the reason and try to arrange a new appointment within the established window period or an unscheduled appointment. In case it is not possible to make an appointment, it will be asked about the presence of adverse events and the reason for leaving the study, such as data.

All materials to be delivered to the subject will be submitted for approval by the corresponding committees.

#### 6.2.5 Identification of the subject.

The study patients will be identified by a number and the initials of their name.

The initials of the subject of study will be obtained starting with the first letter of the name, followed by the first letter of the first surname and the first letter of the second surname, obtaining maximum three letters, in case the person has two names or last name always composed the first letter will be used

#### Example:

- 1. Arieh Daniel Mercado Carrizalez
  - a. Initials: AMC
- 2. Juan De la Torre Orozco
  - a. Ilnitials: JDO

At the counting stage, the participant number will be assigned consecutively, using 3 consecutive digits. Once the subject has been selected, he will be assigned a number with which he will be identified throughout the study. Said code will be composed of eight numbers in the following order from left to right:

- Three digits of the molecule under study according to the denomination by the sponsor.
- Two digits corresponding to the research center number.
- Three digits of the number consecutive to their inclusion assigned in the research center.

#### Example:



#### 6.3 Intervention.

The subjects will be divided into two equal groups, to which they will be assigned randomly and blinded to one of the products under investigation (PI) PRO-122 or Krytantek Ofteno<sup>®</sup>.

Dosage: 1 drop every 12 hours, in both eyes.

<u>Instructions for administration:</u> instillate a drop in the conjunctival sac, it is recommended to exert gentle traction on the lower eyelid, with the index finger, to expose the cul-de-sac and instillation. Avoid blinking energetically for the next few minutes or closing your eyes forcefully.

<u>Duration of the intervention:</u> 7 days.

#### 6.3.1 Medications administered.

#### 6.3.1.1 Drug under study.

#### - PRO-122

- Active ingredients: Timolol 5 mg / ml, brimonidine 2 mg / ml and dorzolamide 20 mg / ml. See Table 6. Quali-quantitative formulation of PRO-122 [32]
- o Pharmaceutical form: Preservative-free ophthalmic solution
- Presentation: multi-dose dropper bottle, 5ml
- Prepared by: Sophia Laboratories, S.A. of C.V.
- Dosage: 1 drop every 12 hours for 7 days, both eyes.
- Description of the solution: clear solution, free of visible particles, with a pH range of 5.4 to 5.9 and a slightly yellow color
- Description of container: White bottle with capacity for 5mL, made of low density polyethylene. Device-closing high density polyethylene assembly, which has a system of silicone and low density polyethylene valves, which allows to keep the sterile solution without the need for additives.

#### *6.3.1.2 Reference treatment.*

#### Krytantek Ofteno®

- Active ingredients: Timolol 5 mg / ml, brimonidine 2 mg / ml and dorzolamide 20 mg / ml See Table 7. Qualitative and quantitative formulation of Krytantek Ofteno® [33]
- Pharmaceutical form: Ophthalmic solution
- o Prepared by: Sophia Laboratories, S.A. of C.V.
- Dosage: 1 drop every 12 hours for 7 days, both eyes
- Description of the solution: clear solution, free of visible particles, with a slightly yellow color.

| Type of agent | Quantity mg/mL | Function |
|---|---|---|
| Dorzolamide hydrochloride | 22.25* | Active principle |
| Timolol Maleate | 6.80 <sup>+</sup> | Active principle |
| Brimonidine tartrate | 2.00 | Active principle |
| Hydroxypropylmethylcellulose | Not showing | Additive |
| Mannitol | Not showing | Additive |
| Citric acid monohydrate | Not showing | Additive |
| Sodium citrate dihydrate | Not showing | Additive |
| Water for the preparation of injectables c.b.p. | 1.00 | Vehicle |

Quali-quantitative formulation of the product under investigation PRO-122. The concentration of the active ingredients is shown, as well as the substances that act as additives.

Table 6. Quali-quantitative formulation of PRO-122.

| Type of agent | Quantity mg/mL | Function |
|---|---|---|
| Dorzolamide hydrochloride | 22.25* | Active principle |
| Timolol Maleate | 6.80 <sup>+</sup> | Active principle |
| Brimonidine tartrate | 2.00 | Active principle |
| Polyethylene glycol monostearate | Not showing | Additive |
| Mannitol | Not showing | Additive |
| Sodium chloride | Not showing | Additive |
| Sodium tetrahydrate decahydrate | Not showing | Additive |
| 50% Benzalkonium Chloride | Not showing | Additive |
| Water for the preparation of injectables c.b.p. | 1.00 | Vehicle |

Quali-quantitative formulation of the investigational drug Krytantek Ofteno® Reg. No. 074M2007 SSA IV. The concentration of the active ingredients is shown, as well as the substances that act as additives.

Table 7. Krytantek Ofteno® qualitative-quantitative formulation.

#### 6.3.2 Strategies to improve adherence and procedure to monitor adherence.

- 1. Direct questioning by the PI about the application of the intervention.
- 2. Delivery of printed chronogram specifying the date of the visit and its activities
- 3. Journal of the subject.

#### 6.3.2.1 Procedure to monitor adherence.

For more than four decades, there have been numerous investigations on the proper way to measure and quantify adherence to medications, nevertheless none has reached consensus to

<sup>(\*)</sup> Equivalent to 20.00 mg / mL of Dorzolamide (+) Equivalent to 5.00 mg / mL of Timolol.

<sup>(\*)</sup> Equivalent to 20.00 mg / mL of Dorzolamide (+) Equivalent to 5.00 mg / mL of Timolol.

PRO-122

establish itself as the gold standard, both in cross-sectional and longitudinal studies. [34] [35] [36] [37] [38] [39] [40] [41]

There are different procedures to measure the adherence of pharmacological interventions. The most common procedure includes self-reports, these include: patient interviews, questionnaires and self-monitoring journals. Its strengths are speed, flexibility, low cost and ease of implementation; they have a high degree of specificity for non-adherence, however, the sensitivity and reliability for adherence is low. [41] [42]

The biochemical measurement of the drug, or its metabolite, is one of the methods that best confirms the use of the drug. However, in addition to raising costs and being impractical, it is of little use in the context of ophthalmic applications, since concentrations at the peripheral level could be undetectable; and samples from other tissues imply more invasive methods that would not be advisable. [41]

Medication counting is another way to measure adherence. Classically referred to as "pill counting", in ophthalmology it is translated to the weight of the bottle. This is a simple, economical and non-invasive method. The main disadvantages of this method are: 1. The application of the medication can not be confirmed (it could have been intentionally thrown or instilled out of the eye) and 2. It depends on the subject bringing back the medication. [41] [42]

For the purposes of this study, the evaluation of the adherence will be favored by means of the diary of the subject, and will be carried out in the following way:

$$Ad = (A_r)100/A_i$$

Ad = Adherence

Ar = Registered applications

Ai = Applications indicated for the intervention

The final adhesion will be determined by the average of the adherence of each one of the visits. Overall adherence (all subjects) will be determined by the average final adherence of each of the subjects.

# 6.3.3 Treatments and concomitant medications allowed and prohibited during the study.

The use of concomitant medications by any route of administration during the intervention period will not be allowed. Except those specified for the study procedures. The objective of this restriction is to avoid pharmacological interactions that could alter the results of the evaluated variables. Nor is the use of herbal or naturist products, whose purpose is to modify some physiological function of the subject.

#### 6.3.4 Treatment management.

The PIs will be provided by Sophia Laboratories, S.A. of C.V. It will be the responsibility of the sponsor to select and ensure the logistic methods for the distribution of the medication. They will be labeled and reconciled. The handling of the treatment will be under the responsibility of the researcher or a designated member of his team.

#### 6.3.4.1 Delivery and reception.

The delivery will be made through a courier service hired by the sponsor, specifically selected for this purpose, at the address of the research center according to the study plan.

PRO-122

Version 1

The reception will be exclusively carried out by the non-blind staff of the research team. You must check the good condition of the primary packaging (box). In case it shows alterations or defects in its integrity that from its judgment could have damaged the content should report it to the sponsor. If the package does not show significant defects, it will proceed to open it.

Inside you must locate the acknowledgment document and the logger (data logger) of temperature and humidity. You should check that the registered temperature and humidity comply with the specifications for transport and shelter (see section 6.3.4.2 Storage). Verify the content (PI) with what is reported in the document. In case the document corresponds to the content, it will sign the receipt and send it to the sponsor. Otherwise, notify the sponsor.

#### 6.3.4.2 Storage.

Storage and safekeeping is the responsibility of the sponsor and the research center. The medication must be stored in a secure area with restricted access.

The storage temperature should be 2 ° to 30 ° C.

The research center has the obligation to record, in the designated format, the temperature recorded in the data logger, every day while the protocol is in force and has PIs.

These data will be compared by the clinical monitor according to the registration in the data logger.

#### 6.3.4.3 Return.

The return will be made by the research center when the sponsor indicates it. Prior to the return, the research center must make a count of the assigned medication and the remaining medication, with the aim of creating an inventory which serves for the final filling of the medication return form.

#### 6.4 Delay variables.

#### 6.4.1 Security variables.

#### 6.4.1.1 Primary outcome variables.

Incidence of adverse events.

#### 6.4.1.2 Variables of primary outcome of tolerability.

- ICO score.

#### 6.4.1.3 Variables of secundary outcome

- Changes in visual ability
- Changes in corneal and conjunctival staining with lysine green.
- Changes in corneal and conjunctival staining with fluorescein.
- Changes conjunctival hyperemia.
- Incidence of chemosis.
- Incidence of alterations in the results of laboratory tests.
- Incidence of alterations in the FC.
- Incidence of alterations in the FR.
- Incidence of alterations in the TAS.

#### 6.4.2 Exploratory variables.

Changes in PIO.

6.4.3 Methods and scales to be used for the measurement of the variables.

| Variable | Kind | Unit<br>(Symbolo) | Method of measurement | Normal<br>value | Evaluation time | Statistical test |
|---|---|---|---|---|---|---|
| Primary | | | | | | |
| Adverse<br>events | Discreet Categorical | Number of cases (n) Present / | Count | 0 | VB, V1, VF y<br>LLS | Mann-<br>Whitney U<br>χ2 or |
| | rating | absent | | Absent | LLS | Fisher's<br>exact |
| ICO score | Discreet | points | Questionnaire | NA | VB, VF | Mann-<br>Whitney U |
| Secondary | | | | | | |
| Visual ability | Discreet | Fraction | Snellen Primer | 1 | VB, V1 y VF | Mann-<br>Whitney U |
| Corneal and conjunctival staining with fluorescein | Ordinal | Degrees | Direct observation<br>with slit lamp and<br>cobalt blue filter,<br>Oxford scale<br>graduation | 0 | VB, V1 y VF | χ2 or<br>Fisher's<br>exact |
| Corneal and conjunctival staining with lysamine green | Ordinal | Degrees | Direct observation<br>with slit lamp,<br>Oxford scale<br>graduation | 0 | VB, V1 y VF | χ2 or<br>Fisher's<br>exact |
| Conjunctival<br>hyperemia | Ordinal | Normal /<br>Very Light /<br>Mild /<br>Moderate /<br>Severe | Direct observation.<br>Classification of<br>Efron. | Normal | VB, V1 y VF | χ2 or<br>Fisher's<br>exact |
| Chemosis | Categorical rating | Present /<br>absent | | Absent | VB, V1 y VF | χ2 or<br>Fisher's<br>exact |
| FC | Discreet | Beats per<br>minute (I /<br>m) | Auscultation with stethoscope | 60 a 100 | VB, V1 y VF | Mann-<br>Whitney U |
| FR | Discreet | Breaths per<br>minute (r /<br>m) | Auscultation with stethoscope | 12 a 24 | VB, V1 y VF | Mann-<br>Whitney U |
| TAS | Discreet | Millimeters<br>of mercury<br>(mmHg) | Measurement with sphygmomanometer | 90-120/<br>60-80 | VB, V1 y VF | Mann-<br>Whitney U |
| Erythrocytes | Continious | Thousands<br>per<br>microliter<br>(Mil / dL) | Laboratory analysis | 4.0- 6.3 | VB y VF | Mann-<br>Whitney U |
| Hemoglobin | Continious | Grams over deciliter (g / dL) | Laboratory analysis | 11.0-16.0 | VB y VF | Mann-<br>Whitney U |

| Variable | Kind | Unit<br>(Symbolo) | Method of measurement | Normal<br>value | Evaluation time | Statistical test |
|---|---|---|---|---|---|---|
| Hematocrit | Continious | Percentage<br>(%) | Laboratory analysis | 36-51 | VB y VF | U de Mann-<br>Whitney |
| VGM | Continious | Femto liters<br>(fL) | Laboratory analysis | 80-97 | VB y VF | U de Mann-<br>Whitney |
| НСМ | Continious | Picograms<br>(pg) | Laboratory analysis | 25-32 | VB y VF | U de Mann-<br>Whitney |
| Leukocytes | Continious | Thousands<br>per liter<br>units (Mil /<br>uL) | Laboratory analysis | 4.0-11.0 | VB y VF | U de Mann-<br>Whitney |
| Platelets | Continious | Thousands<br>per liter<br>units (Mil /<br>uL) | Laboratory analysis | 150-400 | VB y VF | U de Mann-<br>Whitney |
| Glucose | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 70-100 | VB y VF | U de Mann-<br>Whitney |
| Urea | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 10-50 | VB y VF | U de Mann-<br>Whitney |
| Creatinine | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0.6-1.1 | VB y VF | U de Mann-<br>Whitney |
| Glutamic<br>pyruvic<br>transaminase | Continious | Units over<br>liter (U / L) | Laboratory analysis | 0-31 | VB y VF | U de Mann-<br>Whitney |
| Oxalacetic glutamic transaminase | Continious | Units over<br>liter (U / L) | Laboratory analysis | 0-32 | VB y VF | U de Mann-<br>Whitney |
| Total<br>bilirubin | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0-1.1 | VB y VF | U de Mann-<br>Whitney |
| Direct<br>bilirubin | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0.0-0.3 | VB y VF | U de Mann-<br>Whitney |
| Indirect<br>Bilirubin | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0.0-0.8 | VB y VF | U de Mann-<br>Whitney |
| Exploratory | | | | | | |
| Intraocular<br>pressure | Continious | Millimeters<br>of mercury<br>(mmHg) | Goldmann<br>Tonometry | 10 to 21 | VB, V1 y VF | U de Mann-<br>Whitney |

Version 1

The following describes the methods and scales that will be used to measure the variables, which are in strict alphabetical order:

#### 6.4.3.1 Visual capacity.

Visual acuity (VA) is a test of visual function. Spatial visual acuity is the ability to distinguish separate elements of an object and identify them as a whole. It is quantified as the minimum separation angle (located at the nodal point of the eye) between two objects that allows perceiving them as separate objects.

The Snellen notation is described as the distance at which the test is performed, divided by the distance at which the letter is vertically equivalent to 5 arc minutes. Thus, at 6 meters a letter 6/6 (20/20) equals 5 minutes of arc, a letter 6/12 (20/40) equals 10 minutes, and a letter 6/60 (20/200) equals 50 minutes The Snellen fraction can also be expressed as a decimal (ie 20/20 = 1 and 20/40 = 0.5). [43]

The VA will be evaluated basally, without refractive correction with the Snellen chart. Which will be located in a place with adequate lighting, natural or artificial and at a distance of 3m from the subject to be evaluated. The visual acuity of each eye will be taken, starting with a right eye (DO) asking the subject to keep both eyes open and using an occluder to cover the left eye (OS); the subject will read aloud the lines that the evaluator points out, the line of smaller letters that he reaches to see will be annotated by the fractional evaluator as the DO of the DO in the clinical file. Proceed to the OS with the same method.

Subsequently the best refractive correction of the subject will be made and the examination will be repeated using the obtained refraction. This result will be reported as CV, it will be written in fraction in the clinical file and in the CRF, in addition in the CRF it will be written in decimal. By definition, the CV can not be inferior to the AV.

#### 6.4.3.2 Comprehensive ophthalmologic evaluation.

It refers to the ophthalmological exploration of eyelids and appendages, anterior segment and posterior segment that is performed in a routine ophthalmologic review, whose procedures are not specifically included in the study variables. This evaluation has the purpose of identifying unexpected events. The evaluation of the posterior segment will be carried out under drug mydriasis (Tropicamide 0.8% / Phenylephrine 5%), in the slit lamp with an aerial loupe (at the choice of the IP). An integral assessment of the fundus (including optic disc, posterior pole and periphery) will be performed in search of abnormalities that alter the result of the study. The result of the assessment will be recorded in the clinical file. In the CRF it will be registered as normal, abnormal or abnormality that does not affect.

#### 6.4.3.3 Eye comfort index.

It is a questionnaire designed to measure the irritation of the ocular surface with Rasch analysis to produce estimates on a linear scale of intervals (ratings: 0-100). Similar to the index for ocular surface diseases, the ocular comfort index (ICO) evaluates symptoms. The ICO contains items that focus on the discomfort associated with alterations of the ocular surface. Each of these questions has two parts, which inquire separately the frequency and severity of the symptoms. [44] See Annex Index of ocular confort

The evaluator will deliver the questionnaire to the subject and allow the subject to answer it calmly without any pressure and / or coercion, will only assist him if he has difficulty understanding any of the questions.

#### 6.4.3.4 Integrity of ocular surface:

This will be done by means of biomicroscopy using the slit lamp of the research center. A full assessment of the previous segment will be made, which will be recorded in the clinical file. The lighting techniques used will be at the discretion of the IP.

The variables that will be registered in this protocol are:

#### - Conjunctival hyperemia.

It is defined as the simplest reaction of the conjunctiva to a stimulus, a red appearance secondary to the vasodilation of the conjunctival vessels of variable intensity. He will graduate using the Efron scale. [45] See annex Efron scale for conjunctival hyperemia

#### - Chemosis.

It is defined as conjunctival edema, the result of an inflammatory reaction. It is qualified as present or absent. The assessor will use a narrow beam of light at 60 ° and will measure if the conjunctiva separates from the sclera by  $\geq 1/3$  of the total palpebral opening or if it exceeds the gray line. [46]

#### 6.4.3.4.1 Stains.

#### • Staining with green lysine.

A drop of topical anesthetic will be instilled in the conjunctival cul-de-sac, then a second drop will be applied to the tip of the green lysine strip and it will be allowed to slide towards the bottom of the sac. It is essential to quickly evaluate the staining, in sequence, first in the OD and then the OS, so that the observed patterns are equally bright. [47] See annex Scale of Oxford

#### • Fluorescein staining.

A drop of topical anesthetic will be instilled in the conjunctival cul-de-sac, then a second drop will be applied to the tip of the fluorescein strip and it will be allowed to slide towards the bottom of the sac. It is essential to quickly evaluate the staining, in sequence, first in the OD and then the OS, so that the observed patterns are equally bright. This valuation will be done with the cobalt blue filter. [47] See annex Scale of Oxford.

#### 6.4.3.5 Presence of adverse events.

The management of the EAs will be done according to what is described in the Adverse Events section

The PI will register in the corresponding section of the CRF the EAs that come to present the subjects of the study in addition to referring it in the clinical file.

#### 6.4.3.6 Intraocular pressure.

Tonometry is the objective measure of IOP, based primarily on the force required to flatten the cornea or the degree of corneal indentation produced by a fixed force. Goldman's tonometry is based on the Imbert-Fick principle. [43] Tonometry will be performed, after instillation of a drop of topical anesthetic (tetracaine 0.5%), with fluorescein and the use of the cobalt blue filter (after evaluation of corneal surface staining). There will be 3 shots, which will be recorded in the clinical file and the average will be registered in the CRF.

#### 6.4.3.7 Vital signs.

The vital signs to be evaluated (FC, FR and TAS) can be measured by an assistant duly indicated in the organization of the center and the delegation of responsibilities, the technique to be used for the FC and FR will be with the count of repetitions in one minute by direct auscultation with stethoscope.
The SBP should be measured with 5 minutes of previous rest, in the left arm. The instrument can be manual or automatic according to the IP. It is necessary that all measurements are equal in circumstances. The PI will register in the note and the CRF.

#### 6.4.3.8 Laboratory tests.

The designated personnel will perform the extraction of the blood sample, through venipuncture. The vein will be chosen at the discretion of the personnel in charge and will perform asepsis of the skin of the area to be punctured prior to the procedure. It will generate the order of the studies of BH, QS and PFH, to be carried out by the clinical laboratory designated by the sponsor. The clinical laboratory will deliver to the PI the results for its assessment and registration. The normal parameters to be considered will be the ranges established by the laboratory, with a lower and superior margin of 20% in a clinically healthy subject, at the discretion of the PI.

#### 6.4.4 Measurement time.

The measurements of the variables of primary and secondary outcome, as well as the activities contemplated in the protocol, will be carried out and evaluated for each visit, according to the following:

#### Basal Visit / Day 0.

Some of these measurements will be taken at the screening visit to complete the eligibility criteria, at the discretion of the PI, they may be taken to complete the baseline visit data.

- 1. Visual ability
- 2. Intraocular pressure.
- 3. Eye comfort index.
- 4. Ocular surface evaluation.
  - a.It includes stains.
- 5. Comprehensive ophthalmic evaluation
- 6. Evaluation of adverse events.
- 7. Vital signs.
- 8. Evaluation of results of laboratory tests....

## Visit 1 / Day 4.

It can be done in a period  $\pm 1$  days in relation to the 4th day of application.

- 1. Visual ability
- 2. Intraocular pressure.
- 3. Eye surface evaluation
  - a. Includes stains
- 4. Comprehensive ophthalmologic evaluation
- 5. Vital signs
- 6. Evaluation of adverse events.

## Final Visit / Day 8.

It can be done in a period + 1 day in relation to day 8 of the start of application, not before day 8 since the 7 days of application would not be fulfilled.

- 1. Visual ability
- 2. Intraocular pressure.
- 3. Eye comfort index
- 4. Eye surface evaluation
  - a. Includes stains
- 5. Comprehensive ophthalmological evaluation
- 6. Vital signs.
- 7. Evaluation of adverse events.

## Security call / Day 14.

It can be done in a period  $\pm 1$  day in relation to the 14th day of the start of application.

- 1. Ask about the presence of an adverse event.
- 2. Evaluation of results of laboratory tests.

## 6.5 Timeline and study diagram.

| Procedures | Scrutiny | VB | V1 | VF | LIS |
|---|---|---|---|---|---|
| Frocedures | D 1 - X <sup>a</sup> | D 0 | D 4 ± 1 | D 8 a + 1 | D 14 ± 1 |
| CI Signature | Х | | | | |
| Clinic history | Χ | | | | |
| Blood sampling | Χ | | | Χ | |
| Urine pregnancy test | Χ | | | Χ | |
| PIO | Χ | X <sup>1</sup> | X | Χ | |
| CV | Χ | $X^1$ | Х | Χ | |
| Ocular surface stains | Χ | X <sup>1</sup> | X | Χ | |
| Comprehensive ophthalmological evaluation | Х | X <sup>1,2</sup> | Х | X <sup>2</sup> | |
| Vital signs | Χ | $X^1$ | Χ | Χ | |
| Eligibility criteria | Χ | $X_p$ | | | |
| EA evaluation | Χ | Χ | Χ | Χ | X |
| Review of laboratory results | | Х | | | X |
| IP Assignment | | Xc | | | |
| MC evaluation | | Χ | Х | Χ | |
| Delivery of the IP and start of intervention | | Х | | | |
| Ocular Comfort Index | | Х | | Χ | |
| Adherence evaluation | | | Χ | Χ | |
| Daily delivery of the subject | | Х | X | | |
| Continuity evaluation of the subject | | | X | | |
| Return / Evaluation of the subject's Journal | | | Х | Х | |
| Return of PI | | | | Χ | |

a The counting visit may be up to 7 days before the baseline, if it exceeds these days the subject can not enter.

Table 8. Activity Schedule.

b These criteria will be completed with the results of the laboratory tests and those obtained during the screening visit. C Indication to start application the next day.

<sup>1</sup> They can be taken from the scrutiny visit, it is the prerogative of the PI to measure them again at the baseline visit. 2 Includes subsequent segment valuation

## 6.5.1 Procedures to be carried out per visit.

The procedures are listed in the order they are suggested, trying to maintain the consistency of the evaluations and, as far as possible, from the least invasive to the most invasive.

#### 6.5.1.1 Scrutiny visit.

- Informed consent signature: refers to the signing of the written informed consent document. Without obtaining informed consent it is not possible to perform any of the study procedures. See 10.4.1 Obtaining.
- General and ophthalmological clinical history: refers to the technical, clinical and legal document in which the patient's health conditions, medical acts and other procedures performed on the patient are recorded chronologically. Includes anthropometric measurements, anamnesis and comprehensive ophthalmological exploration to discern the patient's eligibility, ie evaluation of both eyes of ocular attachments, exploration with slit lamp of the ocular surface and the anterior segment and fundscopy. If the patient is taken from the established population base of the study center, he / she will be able to use the existing clinical history, and should only perform an update.
- Urine pregnancy test: Refers to the performance of a rapid pregnancy test in all women of childbearing age who wish to enter the study. By fertile age we understand women who have presented their menarche and have not presented their menopause. Menopause is defined as 12 months from the last menstruation in women over 40 years of age; or who have had a bilateral hysterectomy or oophorectomy. Women of childbearing age with contraceptive methods including bilateral tubal obstruction should be tested for pregnancy. This test will be done by the PI or the designated team person according to the instructions of the device delivered by the sponsor.
- Vital signs: see 6.4.3.7 Vital signs.
- Visual capacity: see 6.4.3.1 Visual capacity.
- Integrity of the ocular surface: see 6.4.3.4 Integrity of ocular surface:
- Intraocular pressure: see 6.4.3.6 Intraocular pressure.
- <u>Comprehensive ophthalmological evaluation:</u> see 6.4.3.2 Comprehensive ophthalmologic evaluation
- Sampling of laboratory samples: see 6.4.3.8 Laboratory tests.
- <u>Eligibility criteria:</u> refers to the review by the IP, where it states that the subject can be included in the study by meeting the inclusion criteria and not meeting the exclusion criteria. See 6.2.1 Selection criteria.
- Adverse events: see 6.4.3.5 Presence of adverse events.
- <u>Evaluation of concomitant medications:</u> refers to the interrogation by the PI to the subject, inquiring about the use of medications.

## 6.5.1.2 Baseline visit.

- Review of laboratory tests: refers to the review and analysis by the PI of the results of the BH, QS and PFH.
- <u>Eligibility criteria</u>: with the results of the laboratory the profile of the subject will end for its inclusion or not.
- <u>Evaluation of variables:</u> The data of the evaluation of the variables listed below can be taken from the scrutiny visit. It is the prerogative of the PI to decide whether to use the information from the screening visit or to repeat the evaluations in this visit.
  - o <u>Intraocular pressure</u>
  - Visual ability
  - o <u>Integrity of the ocular Surface</u>

- o Comprehensive ophthalmological evaluation
- o Vital Signs.
- Eye comfort index: see 6.4.3.3.
- Assignment of PI: Refers to determine the intervention that the patient will follow during the study. It will be done according to the Methods section. Assignment of the intervention. This assignment will be made at the baseline visit (day 0) and will go along with the indication to start the treatment period the next day (day 1).
- <u>Delivery of PI:</u> Refers to the delivery of the product under investigation to the patient of the study, by the research center. It will be done according to section 6.3.4.1 Delivery and reception.
- Delivery of the subject's diary: It refers to the delivery by the PI to the subject of the instrument: the subject's diary. The assigned personnel will perform a training on the subject, on the filling of the instrument.
- Adverse events: see 6.4.3.5 Presence of adverse events.
- Evaluation of concomitant medications: See

#### 6.5.1.3 Visit 1

- Return / evaluation of the subject's diary: refers to the submission of the subject's diary to
  the PI by the subject. The PI will review the journal to assess its correct filling, and the
  registration of the applications.
- Adherence evaluation: refers to the assessment performed by the PI according to the section Procedure to monitor adherence.
- Delivery of the subject's diary: see Basal visit.
- Adverse events: see 6.4.3.5 Presence of adverse events.
- Vital signs: see 6.4.3.7 Vital signs.
- Visual capacity: see 6.4.3.1 Visual capacity.
- <u>Integrity of the ocular surface:</u> see 6.4.3.4 Integrity of ocular surface:
- Intraocular pressure: see 6.4.3.6 Intraocular pressure.
- Evaluation of concomitant medications: See 6.5.1.1
- <u>Continuity assessment of the subject:</u> refers to the determination by the PI and desire of the subject to continue with their participation in the study.

#### 6.5.1.4 Final visit

- 6.5.1.5 Return of the IP: refers to the return by the subject, of the surplus IP, to the center.
- 6.5.1.6 Return / evaluation of the subject's diary: see Visit 1.
- 6.5.1.7 <u>Adherence evaluation:</u> refers to the assessment made by the PI according to section 6.3.2.1 Procedure to monitor adherence.
- 6.5.1.8 Adverse events: see 6.4.3.5 Presence of adverse events.
- 6.5.1.9 Urine pregnancy test: see Screening visit.
- 6.5.1.10 <u>Vital signs:</u> see 6.4.3.7 Vital sign<u>s.</u>
- 6.5.1.11 Visual capacity: see 6.4.3.1 Visual capacity.
- 6.5.1.12 <u>Comprehensive ophthalmological evaluation:</u> see 6.4.3.2. Comprehensive ophthalmological evaluation
- 6.5.1.13 Integrity of the ocular surface: see 6.4.3.4 Integrity of ocular surface:
- 6.5.1.14 <u>Intraocular pressure</u>: see 6.4.3.6 Intraocular pressure.
- 6.5.1.15 <u>Sampling of laboratory samples:</u> see 6.4.3.8 Laboratory tests.
- 6.5.1.16 Eye comfort index: see 6.4.3.3 Eye comfort index
- 6.5.1.17 <u>Evaluation of concomitant medications:</u> See ****

## 6.5.1.18 Security call.

- Adverse events: see 6.4.3.5 Presence of adverse events.
- Review of laboratory tests: see Baseline visit.

#### 6.5.1.19 Early termination visit.

If the research subject's participation ends earlier than scheduled, due to an adverse event or any other situation, an unscheduled visit will be made, which will serve as the final visit. In case the subject refuses to attend, the last visit made will be taken as final. Subsequently, the security call will be made in the normal time established.

## 6.5.2 Study diagram.

The diagram of the study contemplates the following:



Figure 3. Diagram of the study.



<sup>\*</sup> Baseline measurements can be taken from those made during the screening visit. It is the investigator's prerogative to perform them again at the baseline visit.

Figure 4. Vertical diagram of the study.

## 6.6 Sample size.

A total size of 24 subjects is estimated, divided into 2 intervention groups. (12 subjects per group). A 45-day enrollment time is expected for the total sample.

## 6.6.1 Calculation of the sample size.

Although there are no references on the calculation of sample size in phase I studies, and the formulation of Krytantek Ofteno® has not reported serious adverse events in its periodic safety reports, it was considered pertinent to be based on the study by Baiza et al (2012). [24]

The sample size was calculated using the formula for proportions

$$n = \left[ (p1)(p2) + (p1)(p2) \left( \frac{Z_{1-\alpha}}{2} + Z_{1-\beta} \right)^2 \right] / (p1 - p2)^2$$

With a statistical confidence of 95% corresponding to the type I error, equal to 1.96, with a power of 80%, corresponding to the type II error, equal 0.84. We considered the presence of 3 adverse events (5.36%), after the use of a triple fixed combination (timolol + brimonidine + dorzolamide) compared to the presence of 5 adverse events (8.93%) of a double fixed combination (timolol, brimonidine) reported in a clinical trial to evaluate efficacy and safety with 112 Mexican subjects with primary open angle glaucoma and / or intraocular hypertension. [24]

According to the previous calculation, the result is 8.12 subjects (8) per group. The total when considering 2 intervention groups is 16 subjects, which was increased by a percentage for the probable losses. The total sample size required is **24 subjects**. Therefore, each group will consist of 12 subjects, who will bring both eyes to the analysis (24 eyes per group).

#### 6.7 Recruitment.

It is essential that, if necessary during the development of this research protocol, the principal investigator requests the approval of the Research Ethics Committee and the Research Committee, as well as the authorization of COFEPRIS, to publish or disseminate in the media. Mass communication, the invitation to participate in the study to those people who meet the selection criteria.

It is possible to discuss with other health professionals the opportunity for healthy subjects to be evaluated by an ophthalmologist at no cost, as well as cabinet exams that will allow the more accurate determination of their ocular clinical status by participating in a sponsored clinical research protocol by Sophia Laboratories, S.A of C.V.

# 7. Methods. Assignment of the intervention

## 7.1 Generation of the allocation sequence.

Two strata corresponding to the intervention groups will be used, which will be balanced for a research center. The allocation will be 1: 1. The generation will be carried out by a third party, authorized by Sophia Laboratories, S.A of C.V., through its electronic system. The information corresponding to this third party will be found in the master folder of the study.

## 7.2 Blinding mechanism.

Blinding will be performed by the Clinical Operations Management of Sophia Laboratories, S.A of C.V. Which will consist in the elimination of the primary label (commercial) in the case of Krytantek Ofteno® and the placement of an identical label to the other interventions. Because the bottle in which Krytantek Ofteno® is packaged differs in the color and shape of the lid used for PRO-122, a masking will be made in the primary packaging which will be identical for the interventions. The subject will be determinedly prohibited from discussing with another person other than the pharmacist aspects related to the vial.

## 7.3 Implementation

The sequence will be generated by means of an electronic randomisation system. Said system will be hired by Sophia Laboratories, S.A of C.V. to a third party. The information corresponding to this third party will be found in the master folder of the study.

## 7.4 Blinding (Masking).

Blinding will correspond to the principal investigator and subinvestigator. In addition, the statistical analysis will be carried out in a blinded manner for the final analysis. Blinding can not be guaranteed in the subject.

The masking will be done through the secondary container. The primary packaging will not be masked by the morphological difference between them. The sponsor and the research center will have two blind / non-blind teams.

They will be identified by means of identical labels. Which, in accordance with current and applicable regulations, must contain at least:

- Name, address and telephone number of the sponsor.
- Pharmaceutical form and route of administration.
- Lot Number.
- Caption "Exclusively for clinical studies"
- Date of Expiry

### 7.4.1 Opening of blinding.

Blinding may be opened in the following cases:

- 1. Presence of a serious adverse event.
- 2. Safety alarm due to the use of the drugs under study.
- 3. In case the sponsor determines it for any reason of security or other reason that considers pertinent.
- 4. In the event that the regulatory authority or the ethics committee so rightly requests so judging it necessary.

# 8. Methods. Collection, administration and data analysis.

### 8.1 Methods of data collection.

Clinical monitors will be assigned, who will be authorized to monitor, review, procure and ensure that the quality of the information obtained from the participants is reliable and trustworthy. Each monitor will schedule periodic visits to the research centers in order to review the source documents and corroborate the information captured in the case report format (CRF). All clinical monitors will be trained in relation to the information of the study protocol (objective, visits, procedures, range of accepted values, etc.). In case the data are not identical between the two registers, the clinical monitor will generate a discrepancy, which must be resolved by the research center at the time that the sponsor deems reasonable to meet the objectives of the clinical study. The correction of the discrepancies will be made according to the Good Documentation Practices.

The data registered in the CRF will be reviewed by personnel of Sophia Laboratories, trained in the ophthalmological, clinical and pharmacological area, which will be able to generate discrepancies in the event that the data do not adhere to the stipulations of the research protocol or put participants at risk.

Once all discrepancies generated by the team of clinical monitors and clinical staff have been resolved, the data will be downloaded into an electronic database (Excel Sheet) by personnel designated by the sponsor. A new revision of the data will be carried out to corroborate the fidelity of the same and new discrepancies may be generated in case it is considered as such.

The database generated will be safeguarded by the sponsor and will only have personal access designated by the same.

## 8.1.1 Strategies to complete the follow-up.

- You will be informed in a clear way the importance of the study and the benefits that the population will obtain from the results of the study.
- Transportation assistance will be provided in order for the participant to attend their visits.
- Calls, messages or a printed calendar will be made in order to remind the participant of their
  appointments and the activities that will be carried out, in addition to the estimated time
  of the same.
- In case the participant does not attend his / her appointment, the research center must make a call to know the reason and try to arrange a new appointment within the established window period or an unscheduled appointment.
- In case it is not possible to make an appointment, it will be asked about the presence of adverse events and the reason for leaving the study, as minimum data.

#### 8.2 Data management.

The subject's medical record (including clinical notes, test results, etc.), as well as the subject's diary, and the ICO questionnaire are considered source data.

The PI or the designated person of your team will fill out the Case Report Format (CRF) as well as all other documents provided by the sponsor (for example, documents related to the handling of the treatment).

An electronic CRF was designed to record the data that are required in the protocol and that the researcher collects in each of the visits. This design is made by a third party, authorized by Sophia Laboratories, S.A of C.V., through its electronic system.

In the case of self-assessment questionnaires, it is not allowed for the principal investigator or person responsible for filling in to modify what was written by the subject of the study.

The data capture in the investigator's site will be done by the investigator or the designated person of his team after performing the Medical File. The researcher or a designated person of your team will be trained in filling the CRF.

All corrections to the CRF data should be made by the investigator or the designated person of your team in accordance with the instructions provided.

To ensure the confidentiality and security of the data, user names and access codes will be used to restrict access to the system only to authorized personnel.

The monitor should ensure that all data has been filled in the CRF. After comparing the data against the source documents, the monitor will ask the researcher to make the correction / clarification using clarifications, so that they are answered and closed as quickly as possible. Once the verification by the monitor is finished, the data will be blocked to avoid modifications.

The Clinical Team of Sophia Laboratories, S.A. of C.V. will do the last medical and scientific review and, if necessary, the data is unblocked if necessary (request for clarification, opening of questions, etc.) and the freezing of the data is confirmed at the end of the study.

## 8.3 Statistical methodology.

#### 8.3.1 Analysis of primary and secondary outcome variables.

The statistical analysis will be carried out by personnel of Sophia Laboratories. The statistical program SPSS version 19.0 (IBM Corporation, Armonk, NY, USA) will be used.

The designated personnel will be blinded to the intervention groups. The coding will be done using consecutive numbers for each intervention group.

The data will be collected and sorted in an excel sheet. Later they will be exported to the platform of the SPSS program. The variables will be categorized according to their nature.

The results of the continuous quantitative variables will be presented in measures of central tendency: mean, standard deviation and ranges. See

| Variable | Kind | Unit<br>(Symbolo) | Method of measurement | Normal<br>value | Evaluation time | Statistical<br>test |
|---|---|---|---|---|---|---|
| Primary | | | | | | |
| Adverse events | Discreet | Number of cases (n) | Count | 0 | VB, V1, VF y | Mann-<br>Whitney U |
| | Categorical rating | Present /<br>absent | Observation | Absent | LLS | χ2 or<br>Fisher's<br>exact |
| ICO score | Discreet | points | Questionnaire | NA | VB, VF | Mann-<br>Whitney U |
| Secondary | | | | | | |

| Variable | Kind | Unit<br>(Symbolo) | Method of measurement | Normal<br>value | Evaluation time | Statistical<br>test |
|---|---|---|---|---|---|---|
| Visual ability | Discreet | Fraction | Snellen Primer | 1 | VB, V1 y VF | Mann-<br>Whitney U |
| Corneal and<br>conjunctival<br>staining<br>with<br>fluorescein | Ordinal | Degrees | Direct observation with slit lamp and cobalt blue filter, Oxford scale graduation | 0 | VB, V1 y<br>VF | χ2 or<br>Fisher's<br>exact |
| Corneal and conjunctival staining with lysamine green | Ordinal | Degrees | Direct<br>observation with<br>slit lamp, Oxford<br>scale graduation | 0 | VB, V1 y<br>VF | χ2 or<br>Fisher's<br>exact |
| Conjunctival<br>hyperemia | Ordinal | Normal /<br>Very Light /<br>Mild /<br>Moderate /<br>Severe | Direct observation.<br>Classification of<br>Efron. | Normal | VB, V1 y VF | χ2 or<br>Fisher's<br>exact |
| Chemosis | Categorical rating | Present /<br>absent | | Absent | VB, V1 y VF | χ2 or<br>Fisher's<br>exact |
| FC | Discreet | Beats per<br>minute (I /<br>m) | Auscultation with stethoscope | 60 a 100 | VB, V1 y VF | Mann-<br>Whitney U |
| FR | Discreet | Breaths per<br>minute (r /<br>m) | Auscultation with stethoscope | 12 a 24 | VB, V1 y VF | Mann-<br>Whitney U |
| TAS | Discreet | Millimeters<br>of mercury<br>(mmHg) | Measurement with sphygmomanometer | 90-120/<br>60-80 | VB, V1 y VF | Mann-<br>Whitney U |
| Erythrocytes | Continious | Thousands<br>per<br>microliter<br>(Mil / dL) | Laboratory<br>analysis | 4.0- 6.3 | VB y VF | Mann-<br>Whitney U |
| Hemoglobin | Continious | Grams over deciliter (g / dL) | Laboratory analysis | 11.0-16.0 | VB y VF | Mann-<br>Whitney U |
| Hematocrit | Continious | Percentage<br>(%) | Laboratory analysis | 36-51 | VB y VF | U de Mann-<br>Whitney |
| VGM | Continious | Femto liters<br>(fL) | Laboratory analysis | 80-97 | VB y VF | U de Mann-<br>Whitney |
| НСМ | Continious | Picograms<br>(pg) | Laboratory analysis | 25-32 | VB y VF | U de Mann-<br>Whitney |
| Leukocytes | Continious | Thousands<br>per liter units<br>(Mil / uL) | Laboratory analysis | 4.0-11.0 | VB y VF | U de Mann-<br>Whitney |

| Variable | Kind | Unit<br>(Symbolo) | Method of measurement | Normal<br>value | Evaluation time | Statistical<br>test |
|---|---|---|---|---|---|---|
| Platelets | Continious | Thousands<br>per liter units<br>(Mil / uL) | Laboratory analysis | 150-400 | VB y VF | U de Mann-<br>Whitney |
| Glucose | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 70-100 | VB y VF | U de Mann-<br>Whitney |
| Urea | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 10-50 | VB y VF | U de Mann-<br>Whitney |
| Creatinine | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0.6-1.1 | VB y VF | U de Mann-<br>Whitney |
| Glutamic<br>pyruvic<br>transaminase | Continious | Units over<br>liter (U / L) | Laboratory analysis | 0-31 | VB y VF | U de Mann-<br>Whitney |
| Oxalacetic glutamic transaminase | Continious | Units over<br>liter (U / L) | Laboratory analysis | 0-32 | VB y VF | U de Mann-<br>Whitney |
| Total<br>bilirubin | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0-1.1 | VB y VF | U de Mann-<br>Whitney |
| Direct<br>bilirubin | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0.0-0.3 | VB y VF | U de Mann-<br>Whitney |
| Indirect<br>Bilirubin | Continious | Milligrams<br>over deciliter<br>(mg / dL) | Laboratory analysis | 0.0-0.8 | VB y VF | U de Mann-<br>Whitney |
| Exploratory | | | | | | |
| Intraocular<br>pressure | Continious | Millimeters<br>of mercury<br>(mmHg) | Goldmann<br>Tonometry | 10 to 21 | VB, V1 y VF | U de Mann-<br>Whitney |

The Kolmogorov-Smirnov test will be performed to determine if the distribution presents normality in the results obtained in each study group [48].

The statistical analysis of the continuous **quantitative variables** to find significant differences (p) will be the following:

- Intra-group analysis: will be determined by the Wilcoxon rank test, for quantitative variables [49]
- <u>Inter-group analysis:</u> Kruskal-Wallis test [50]. This non-parametric test will be used to test whether a group of data comes from the same population. Intuitively, it is identical to the

ANOVA with the data replaced by categories. For the quantitative variables, the student's t-statistic will be used.

The level of difference to consider significance will be an alpha of 0.05 or less.

The result of nominal and ordinal qualitative variables will be presented in frequencies, proportions and percentages. See table 1 (section 6.4.3).

The statistical analysis to identify significant differences of the qualitative variables will be done creating 2x2 contingency tables and it will be done in the following way:

- <u>Intra-group difference:</u> McNemar test [51]. Which is applied to 2 × 2 contingency tables with a dichotomous trait, with pairs of matched subjects, to determine if the marginal frequencies of row and column are equal (marginal homogeneity).
- <u>Inter-group difference:</u> Pearson's χ2 test (or Fisher's exact).

The level of difference to consider significance will be an alpha of 0.05 or less.

For the reporting of adverse events all eyes of those participants who were randomly assigned to an intervention group after the baseline visit will be considered. The results will be expressed in number of cases (eyes).

The final report of the results will be shown in tables or graphs, as appropriate.

It will be considered that the investigational drug is safe and tolerable when there are no clinical and statistical differences in all the variables of primary outcome, with respect to its comparators.

Those subjects who comply with an adherence greater than 60% will be included in the statistical analysis to meet the objective of the study, taken from the subject's diary. It was considered that from the minimum dose necessary to obtain a pharmacological effect (hypotensive / 1 application per day) and the presence of adverse events (exposure) is sufficient to meet the overall design objective, according to the pharmacological characteristics of the product in investigation.

#### 8.3.2 Additional analyzes.

No additional analyzes are contemplated to those previously described. However, these may be performed if during the conduction of the study it is required to analyze specific safety aspects of any intervention, maintaining the blinding until the end of the study.

#### 8.3.3 Population analysis and management of missing data.

An intention-to-treat analysis will be carried out, where the data of the participants who have completed the Visit 1 will be included.

# 9. Methods. Monitoring.

## 9.1 Data monitoring.

Monitoring visits by a monitor from Laboratorios Sophia, S.A. of C.V. are intended to confirm that the studies sponsored by Sophia Laboratories, S.A. of C.V. they are conducted in accordance with

the ethical principles that have their origin in the Declaration of Helsinki and that are consistent with the Good Clinical Practices and with the applicable regulatory requirements.

The researcher must ensure that they have sufficient time, space and qualified personnel for the monitoring visits.

Sophia Laboratories, S.A. of C.V. will monitor the study to verify, among other things, that:

- The data is authentic, correct and complete.
- They are protecting the security and rights of the subjects.
- The study is being carried out in accordance with the currently approved protocol, any other study agreement, Good Clinical Practices and all applicable regulatory requirements.

The details of the monitoring are documented in the Monitoring Plan (PM). The PM describes: the frequency and level of detail with which the monitoring will be performed, the activities to be carried out during the study according to its role (blind / non-blinded), the description of deviations from the protocol and its management.

#### 9.2 Adverse events.

Perform the verification of adverse events through questioning, review of the information recorded in the journal of the subject, relevant physical examination, assessment of evolution, as well as the appropriate medical and pharmacological management, resolution or outcome and final discharge following the definitions determined in the national and international regulations. [67] [68] [69]

In the event of adverse events or any event that puts the health and well-being of patients at risk, appropriate medical attention will be provided, either at the research site or referred to the Hospital Center with the greatest resolving power researcher and / or researcher site have medical care agreement. The researcher will notify the clinical monitor of the sponsor, according to the times established in the national and international regulations. In the case of serious adverse events, notify the sponsor and record the corresponding information in the case report form and in turn inform the Committee of Research Ethics, the Research Committee.

The attention of the adverse events will be made according to the diagram of attention of the event (see Figure 5. Attention of the adverse event).

In the final report that will be drafted by the Clinical Team of the Department of Clinical Operations of Sophia Laboratories, S.A. of C.V., will include the report of adverse events in compliance with current national and international regulations. [68] [67]

If the research subject debuted during his participation in the study with an adverse event of a chronic course, such as diabetes or systemic arterial hypertension, he / she will be referred to the competent health professional for chronic treatment and we will adhere to the stipulations of the ICH for monitoring and ending their participation.

### 9.2.1.1 Record of adverse events in the Case Report Form.

The registry of adverse events considers the information about the identification data of the patient involved as code, age, sex, left eye and right eye.

Information about the type of event that is adverse to the IP or to the study medication, as appropriate. The date on which the adverse event occurs is reported, as well as in which the Investigator is aware of it, date of resolution or outcome, as applicable. The clinical diagnosis is indicated. If a lack of therapeutic response to the IP and / or investigational medication is detected,

/ersion 1

it must be reported as a serious adverse event within the period stipulated by current regulations. To include in concomitant medications the therapy used for the pharmacological management of the adverse event. Record the outcome or resolution of the event: patient recovered without sequelae, with sequelae, not recovered. Patient who presented death due to the adverse event, patient who presented death and it is judged that the drug could have contributed, patient who presented death and this is not related to the investigational product or medication, or indicate that it is not known what the consequence of the event is.

Consign information about the product or drug under investigation or the drug associated with the adverse event, adverse reaction or suspected adverse reaction. As applicable, the information concerning generic name, distinctive denomination or code of the IP and / or investigational drug should be recorded, as appropriate according to the methodological design of the study, this is relevant in the case of blinded studies or those where placebo is used as comparators, since there are circumstances that justify opening the cecum to determine if the adverse event may be attributable to the active agent, the combination of active agents, or the pharmacologically inert substance (s), such as the vehicle or additives, as appropriate the clinical research phase in which the development of the drug is located. It will also be necessary to record the data concerning the batch number, manufacturer laboratory, expiration date, dosage, route of administration, start and end dates of administration and / or consumption, reason for the prescription; according to whether it is a product or drug under investigation (protocol in which the patient currently participates) or is a medicine that the subject in question consumes for the treatment of basic concomitant diseases or used for the management of any sign or transient symptom that does not correspond to the Natural History of the pathology that motivated its entry into the research protocol.

Record the withdrawal or maintenance of the medication, IP or investigational medication, as appropriate. Indicate if the adverse event disappears when the IP or investigational medication or suspicious medication is removed (to provoke the event). Also indicate if a dose adjustment is made, if the event changes in terms of intensity or seriousness, persistence of the reaction. It is important to indicate that in those patients who are exposed again to the PI, investigational medication or medication, which had previously been suspended, if the adverse reaction or adverse event reappears.

Regarding concomitant pharmacotherapy. Indicate the generic name, the dose, the route of administration, start and end dates of its use, as well as the reason for the prescription regardless if it is consistent with the information to prescribe or technical data sheet or is used outside the regulations or of what the local, national or international regulatory entity has authorized.

Concerning the relevant clinical antecedents. The analysis of the adverse event considers the information previously reported, notwithstanding the clinical context in which this harmful phenomenon occurs in the participants of the clinical research protocol, it is of special interest, so that information about the previous conditions, phenomena of hypersensitivity or allergy, previous surgical procedures, laboratory analysis or cabinet examinations that have been practiced on the participant, etc., that the investigator deems fit to mention may do so. If you have enough space in the case report format, you can complete the information in your clinical note in the clinical file.

#### 9.2.1.2 Follow-up of adverse events.

The PI will provide the attention and guidance of the EA that the participant presents until the outcome of the same, according to what is referred to the following section.

#### 9.2.1.3 Procedures for a serious adverse event.

The process of attention of the adverse event considers the following stages:



#### Attention to the adverse event.

- 1. During the development and conduct of the present clinical investigation, undesirable damaging events or adverse reactions, of medical involvement, which do not necessarily have a causal relationship with the IP or investigational medication, may occur in the participant patient. These harmful phenomena can occur during the use of investigational drugs, unintentionally, at doses authorized for use in humans; by a local, national or international regulatory entity, whether for prophylaxis, diagnosis, treatment or for the modification of some physiological process. However, it can be suspected that the IP or the investigational drug or the placebo cause some unwanted clinical manifestation. Adverse events, adverse reactions or suspected adverse reactions to one or several medications can occur during the systematic evaluation of the participants (on the days when the clinical review is scheduled, according to the schedule of activities) or suddenly, as such way that;
- 2. The investigator must be the first person to whom the patient reports that they have developed or presented a harmful clinical phenomenon during their participation in this research protocol.

- 3. According to your clinical judgment; on the basis of the pertinent physical examination, questioning, etc., as well as the analysis of the information available in the medical literature and of what is referred to in the researcher's manual, information to prescribe or technical record of the comparator drug, the principal investigator determines the relevant attention of the event / harmful reaction; either,
- 4. At the research site or at the hospital with the greatest resolving power (1st, 2nd or 3rd level of medical attention). In such a way that, in case the patient is sent by the Investigator to a hospital, he / she attends by means of a reference system, it can be with an identification card that the patient belongs to the present investigation and there is an official number or folio, which pertains to the emergency care agreement with the health institution with the greatest resolving power, or a medical reference note issued by the principal investigator, so that appropriate attention is given to the participating patient. It should be noted that the Study Sponsor, Sophia Laboratories, S.A. of C.V., will pay the expenses for the medical attention of the participant patient, only if the adverse event is associated or is in relation to the IP or investigational medication.
- 5. Taking the collected clinical information, either during the care provided in the research site or provided by the treating physician (s) in the hospital, the principal investigator records the adverse event in his / her clinical note of the file clinical setting, indicating the seriousness, intensity (mild, moderate or severe), relationship with the investigational product or drug, as well as,
- 6. The migration of the relevant data to the case report format and to its respective adverse event section; noting the pertinent information, already referred to in section 9.3.1.1., in virtue of the fact that in cases of serious adverse events, which must be notified in less than 24 hours after the moment in which the principal investigator has knowledge of the same, the clinical monitor of the study is informed, so that in turn it informs the Clinical Team and the Pharmacovigilance Department of the sponsor and later it is informed to the Committee of Ethics in Research. With respect to non-serious adverse events, these will be recorded and adequately addressed and the corresponding regulatory entity will be informed about the safety profile of the IP or investigational medication in the final report of the clinical trial.

The record of the outcome of the adverse event depends substantially on the follow-up that the principal investigator makes to the participant, since it is expected that the majority of harmful phenomena, consult section of the safety profile in number 5.3 and in the researcher's manual, are of a nature ophthalmic, however, there may be systemic alterations. Therefore, in the opinion of the researcher, the withdrawal of the participant or his / her permanence will be considered, according to what is stipulated in section 6.2.1.2 Exclusion criteria of the present research protocol.

#### 9.2.1.4 Causality assessment.

The assessment of causality, the methodology used to estimate the probability of attributing a drug, investigational drug or IP to the observed adverse event, considers probabilistic categories, according to the available evidence and the quality of the information, based on the national pharmacovigilance regulations. [67] As a tool to facilitate the probabilistic categorization of causality, the department of pharmacovigilance and tegno-vigilance of Laboratorios Sophia (UFTLS) can use the algorithm of Karch and Lasagna modified by Naranjo referred to by Aramendi I, 2011 in

which different items are scored which allow to assign a value to the cause-effect relationship between the administration of the drug and the adverse reaction. [70] **See Table 9. Algorithm of Karch and Lasagna modified by Naranjo**.

| Num | Reagent | | |
|---|---|---|---|
| ber | neagent | Yes | No |
| 1. | There are previous conclusive reports about the adverse drug reaction, adverse event or suspected adverse drug reaction | +1 | 0 |
| 2. | The adverse event appeared when the suspected drug was administered | +2 | -1 |
| 3. | Adverse reaction to medication, adverse event or suspected adverse reaction to medication improved upon discontinuation or administration of a specific antagonist | +1 | 0 |
| 4. | Adverse reaction to medication / adverse event / suspected adverse drug reaction reappeared when administering the drug / investigational product / investigational medication | +2 | -1 |
| 5. | There are alternative causes that may cause this reaction | -1 | +2 |
| 6. | Adverse reaction / adverse event / suspected adverse drug reaction occurred after placebo administration | -1 | +1 |
| 7. | The drug was determined in blood or other liquids in toxic concentrations | +1 | 0 |
| 8. | The intensity of the adverse reaction / adverse event / suspected adverse drug reaction was higher at higher doses or lower at lower doses | +1 | 0 |
| 9. | The patient has had similar reactions with the drug / product under investigation or investigational medication, in the past | +1 | 0 |
| 10. | Adverse reaction / adverse event / suspected adverse reaction to medication was confirmed with some objective evidence | +1 | 0 |
| | Total score | summ | ation |
| | Probabilistic category based on the score obtained | | |
| I | The causal relationship is checked | ≥,9 | |
| II | It is likely that the RAM is due to the drug or product under investigation | 5 a 8 | |
| Ш | It is possible that the RAM is due to the drug or product under investigation | 1 a 4 | |

Each reagent receives a defined score and the final summation allows estimating the probabilistic category of the cause-effect relationship between the administration of the product under investigation and the adverse reaction, adverse event or suspected adverse reaction.

#### Algorithm of Karch and Lasagna modified by Naranjo.

In such a way that the degree of certainty to establish the IP or investigational medication (as appropriate) as the causal agent of the harmful phenomenon that happens to the participating patient, can be indicated directly by the principal investigator based on his clinical experience or through the voluntary application of the tool mentioned previously. Notwithstanding, it is important that the researcher and the UFTLS take into account the following arguments in favor of the causal relationship:

- a) Strength of association that refers to the number of cases in relation to those exposed.
- b) The consistency of the data, ie the presence of a common characteristic or pattern.
- c) The exposure-effect pattern: which determines the relationship with the site of onset, time, dose and reversibility after suppression.

- d) The biological plausibility: that refers to the possible pharmacological or physiopathological mechanisms involved in the development or presentation of the adverse event.
- e) Experimental findings: for example, the appearance of abnormal metabolites or high levels of drug or the product of its biotransformation.
- f) Analogy: experience acquired with other related drugs, adverse reactions frequently produced by the same family of pharmacological agents.
- g) Nature and characteristics of the data: objectivity, accuracy and validity of the relevant documentation. [71]

## 9.2.2 Responsibilities of the sponsor.

The sponsor will be responsible, and will cover the expenses derived from the medical attention to adverse events related to the IP.

## 9.3 Unanticipated problems.

The unanticipated problems (NAP) consider those situations that pose risks for the participating subjects, in general, any incident, experience or result that meets all the following criteria:

- Unexpected in terms of its nature, severity or frequency in relation to: 1) documents related to the study such as the researcher's manual, study protocol and informed consent format; and 2) the characteristics of the population being studied.
- Related or possibly related to your participation in the study (possibly related means that there
  is a reasonable possibility that the incident, or results, was caused by the study's own
  procedures).
- Indicative that the research places the participants at a higher risk of harm (including physical, psychological, economic or social) than previously recognized.

#### 9.3.1 Report of PNAs.

The PI will be responsible for reporting PNAs to the sponsor, to the CI, to the CEI. The report must contain the following information:

- Identification of the study: protocol title and number, name of the PI and, where appropriate, the center.
- Detailed description of the event, incident, experience or result.
- Explanation, justification of the reasons why the incident represents an NAP.
- Description of changes to the protocol or corrective actions taken or proposed in response to the NAP.

The PNAs that are EAS must be reported to the CEI and the sponsor within the first 24 hours that the PI has knowledge of this.

Any other NAP will be reported to the CEI and the sponsor within the first 5 business days, after the PI has knowledge of this.

### 9.4 Audit.

To guarantee compliance with the PCBs and with all applicable regulatory requirements, Sophia Laboratories, S.A. of C.V. could carry out an audit of quality assurance. Regulatory agencies could also conduct a regulatory inspection of this study.

#### 9.4.1 Pre-study audit.

The study centers included in the study will be subject to a feasibility visit prior to the selection of the center, where it will be verified that they meet the minimum requirements indicated by the sponsor.

#### 9.4.2 Audit / Inspection during the conduction of the study.

They may take place at any time before, during or after the conclusion of the study. If an audit or inspection is conducted, the investigator and the institution must agree to allow the auditor / inspector direct access to all relevant documents, and will allocate their time and that of their staff to the auditor / inspector to discuss the findings and any relevant problems. In case the audit has not been scheduled by the sponsor, the center must notify Sophia Laboratories, S.A. of C.V. immediately.

## 10. Ethical considerations.

## 10.1 Approval of the committees.

The present study will be conducted according to the standards of the Declaration of Helsinki, World Medical Association 2013. Nuremberg Code; Nuremberg Trial by the International Tribunal of Nuremberg, 1947. Belmont Report, National Commission for the Protection of Subjects of Biomedical Research and Conduct, 1979. Will be conducted in accordance with scientific and technical requirements for the registration of medicines for use of the International Conference on Harmonization (The International Council for Harmonization, ICH) Guide to Good Clinical Practices.

International Ethical Guidelines for Biomedical Research in Human Beings of the Council for International Organizations of Medical Sciences (Council for International Organizations of Medical Sciences, CIOMS, 2002). International Ethical Guidelines for epidemiological studies of the Council for International Organizations of Medical Sciences (Council for International Organizations of Medical Sciences, CIOMS, 2008). The Research Ethics Committee and the Research Committee will evaluate the protocol before conducting the study and will issue their approval or possible modifications for its realization, these Committees should be notified of any significant changes to the protocol. In addition to the above, the current regulations issued by the Ministry of Health will also be complied with. General Health Law, NOM 012 Official Mexican Standard NOM-012-SSA3-2012, Which establishes the criteria for the execution of research projects for human health. The study is considered as an investigation with a risk greater than the minimum according to the Regulation of the General Health Law on Health Research, Title Two, Chapter I, Article 17, Category III, published in the Official Gazette on 6 January 1987.

Principal investigators or study coordinators or personnel authorized by the sponsor will be evaluated by the Research Ethics Committees, Research Committees, and when applying to the Biosafety Committee the essential documentation of the research project: research protocol, letter of informed consent, researcher's manual, subject's diary, as well as those requested, in addition, according to local, national or international requirements applicable by regulatory entities.

The study will not start in the research site if you do not have the confidentiality agreements and economic proposal of each of the principal investigators, duly signed and without having previously obtained the favorable opinion and / or the approval of the Committees of Ethics in Research, Research Committees, and when applicable by the Biosafety Committee, corresponding.

The study will not begin without having met the relevant local, national or international regulatory requirements and without having the corresponding health authorization.

## 10.2 Amendments to the protocol.

The amendment procedure will be relevant when there is a need to make any change to a document that is part of the research project or protocol, derived from variations in the <u>methodological structure</u>, substitution of the principal investigator or when identifying risks in the research subjects. The documents subject to amendment will be: protocol, letter of informed consent, researcher's manual, documents for the patient, scales of measurement and schedule of activities.

Any amendment must be approved by the sponsor and / or the principal investigator, the amended document (s), once reviewed and approved by the Research Ethics Committee and the Investigation Committee or when applicable, by the Board of Directors. Biosafety, (entities that issued the initial favorable opinion for the conduct of the investigation) will be sent (s) for authorization by the relevant regulatory entity.

Amendments that substantially modify the protocol, confers an additional or different risk on the research subjects, must be approved by the aforementioned Committees. It is the investigator's responsibility to take action in situations that require immediate action to avoid unnecessary harm to study participants.

The principal investigator has the responsibility to inform the Research Ethics Committee of any amendment to the protocol that could eventually affect the rights, safety or welfare of the research participants. Likewise, he must know any situation or new knowledge that will show a greater risk for the participants, the termination or premature suspension of the study, the reasons and the results obtained up to that moment. You must also inform about the conclusion of the study, when completing the research protocol.

The list of amendments, and in the necessary cases, the relation of the issuance of errata, will be referred to in the final report of the investigation.

## 10.3 Early termination of the study.

The study may be temporarily suspended or terminated prematurely if there is a sufficiently reasonable cause. The written notice, which documents the reason for the suspension or early termination, must be delivered by the executing party of the suspension. The PI must inform the study participants, the CI and the CEI as soon as possible, providing the reasons.

The situations in which the suspension or early termination of the study will be considered include, but are not limited to:

- 1. Presence of serious adverse events in more than 10% of the participants in each intervention group.
- 2. The competent authority (COFEPRIS) considered it for security alerts.
- 3. The Sponsor determined it for your convenience or eventualities such as: economic support, manufacturing errors, etc.
- 4. Less recruitment than stipulated.
- 5. Determination of unexpected risks for participants, which are significant or unacceptable.
- 6. Obtaining new relevant safety information.
- 7. Insufficient adherence to protocol requirements.
- 8. The data obtained are not evaluable or are not sufficiently complete.
- 9. Determination that the primary objective has been reached.
- 10. Determination of futility.

In case of suspension, the study can be resumed once the situations that led to suspension have been remedied; as long as this justification is sufficient for the sponsor, CI, CEI and regulatory authorities.

#### 10.4 Consent.

#### 10.4.1 Obtaining.

The informed consent must be obtained before the subject undergoes any procedure indicated in the protocol.

The written consent documents will incorporate the elements of informed consent described in the Declaration of Helsinki and the ICH Guide to Good Clinical Practices and will be in compliance with all applicable laws and regulations.

The PI will provide the potential participant with all the information regarding the characteristics of the study, its potential benefits, risks, objectives and procedures thereof.

This information will be with a language understandable to the subject, it will be explained to the subject that has the right to interrupt their participation in the study at any stage, without affecting

the relationship with the researcher and / or future assistance. The informed consent will be put to the consideration of the possible participant; this must have enough time to analyze each and every one of the aspects mentioned above and if there is any doubt this will be clarified by the person in charge of obtaining the informed consent.

Once the participant agrees to participate in the study, he / she must sign and date the letter of informed consent in the presence of two witnesses who have or are not related to the subject of the study, who will participate during the informed consent process and will sign endorse that the process was carried out prior to any study procedure, that the study information was clearly explained and doubts were clarified in case of existing.

If a subject is illiterate, the acceptance will be with their fingerprint, and in the event that the subject is not able to grant an informed written consent, a representative of the subject "legally authorized" can provide such consent, the subject in accordance with the applicable laws and regulations.

The PI must also sign and date this consent.

The informed consent must be signed in duplicate by all involved, and two witnesses, one copy will be filed in the researcher's folder and the other will be delivered to the participant. The PI or delegated personnel, must document the process of obtaining the Informed Consent by means of a detailed medical note, where the signed version is specified, the date on which the document was signed and how the process was carried out.

## 10.4.2 Special considerations.

The auxiliary studies that will be carried out during the conduction of the study (laboratory tests) do not pose an additional risk that should be considered apart from the procedures listed in the informed consent.

#### 10.4.3 Modification to informed consent.

Any change to "informed consent" constitutes an amendment to this document and must be presented for approval before the Ethics in Research Committees, and if applicable before the Competent Authorities.

The amendment will include a copy of the new version in the language or languages of the country.

Such amendments may be implemented only after having obtained the written approval of the Research Ethics Committee and the Regulatory Entity (as applicable), with the exception of an amendment that is required to eliminate an immediate danger for the subjects of the study.

Each subject affected by the amendment must complete, date and sign two originals of the new version. The subject will be given a signed original of the amendment and the researcher will keep the second original.

In the event that new information may arise that may be relevant to the subject's decision to continue participating in the study, this information should be communicated in a timely manner to the latter. This information will be provided through an amendment to the informed consent, which must be completed, dated and signed in duplicate through a process of re-consent.

## 10.5 Confidentiality.

All documents and information provided to the researcher by the sponsor are strictly confidential. The researcher expressly agrees that the data on their professional and clinical experience, provided

to the sponsor on paper and stored in electronic format, are only for use related to their activities with the sponsor of clinical studies, in accordance with Good Clinical Practices. The researcher accepts that he / she and the members of his team will use the information only within the framework of this study, to carry out the protocol. This agreement is mandatory as long as the confidential information has not been disclosed to the public by the sponsor. The protocol of the clinical study provided to the researcher may be used by him and by his colleagues to obtain the informed consent of the subjects for the study. The clinical trial protocol, like any information taken from it, should not be disclosed to other parties without the written authorization of the sponsor.

The researcher will not disclose any information without the prior written consent of Sophia Laboratories, S.A. of C.V., except to the representatives of the Competent Authorities, and only by request of the same. In the latter case, the researcher undertakes to inform Sophia Laboratories, S.A. of C.V. before revealing the information to these authorities.

The researcher will fill out and maintain a record of the subjects' selection as well as the identification and enrollment list of each of the subjects participating in the study. The researcher agrees to give on-site access to the auditor and / or the representatives of the Competent Authorities. The information will be treated in compliance with professional secrecy.

## 10.6 Conflict of interests.

The independence of the conduction of the study and its results, of any current or perceived external influence is critical. For this reason, any current conflict of interest of any person who exercises a role in the design, conduct, analysis, publication or any aspect of this study will be declared. Moreover, those people who have a perceived conflict of interest will be asked to handle it in a way appropriate to their participation in the study.

#### 10.6.1 Declaration of interests.

The PI commits to make a declaration of financial interests, as well as a conflict of interests prior to the start of the study.

### 10.7 Access to information.

The final database of the study will be owned by Sophia Laboratories, S.A. of C.V. and your access will be restricted. The PI will not have access to it, unless it has prior written authorization from the sponsor.

## 10.8 Auxiliary care and after the end of the study.

Once the study is finished and the adverse events are closed according to the adverse events section, the sponsor will not extend care on the research subject.

## 10.9 Biosecurity aspects.

#### WITHOUT BIOSECURITY IMPLICATIONS

The present protocol, entitled: "Phase I clinical study, to evaluate the safety and tolerability of the preservative-free ophthalmic solution PRO-122 compared with Krytantek Ofteno®, prepared by Sophia Laboratories, S.A. of C.V. on the ocular surface of ophthalmological and clinically healthy subjects ", and number: SOPH122-0518 / I DOES NOT HAVE BIOSECURITY IMPLICATIONS, since NO

infectious-contagious biological material will be used; pathogenic strains of bacteria or parasites; viruses of any kind; radioactive material of any kind; animals and / or cells and / or genetically modified plants; toxic, dangerous or explosive substances; Any other material that endangers the health or physical integrity of the research center's personnel or the research subjects or affects the environment. It is also stated that cell, tissue or organ transplant procedures or cell therapy procedures will not be carried out in this project, nor will laboratory, farm or wildlife animals be used.

## 10.10 Final report and publication of results.

### 10.10.1 Final report.

Once the statistical analysis is finished, a final report will be drafted with the results obtained, in charge of the Scientific Committee of the Clinical Operations Department of Sophia Laboratories, S.A. of C.V. Said report will be prepared following the recommendations of the E3 Step 4 Guide of the ICH.

#### 10.10.2 Communication of results.

Regardless of the results in the study, Sophia Laboratories, S.A. of C.V., is committed to communicate to the principal investigators and to the corresponding regulatory entities of the countries with participating research centers, the final report of the study. These results will also be shared with the research committee and the CEI. The communication to the research subjects will be the responsibility of the PI. Maintaining at all times the rights on the publication and dissemination of the information contained.

#### 10.10.3 Publication of results.

Sophia Laboratories, S.A. of C.V., acting as the sponsor of the study, assumes full responsibility for its function and retains the exclusive property rights over the results of the study, which may be used in the manner it deems appropriate.

The PI undertakes not to publish or communicate data collected only in a center or in part of the centers before the publication of the full results of the study, unless prior written agreement is given by Sophia Laboratories, S.A. of C.V.

Any publication and / or communication project related to the study and / or the results obtained during the study or after the completion of the study will be presented to participating medical researchers at least 30 days in the case of a publication and 15 days in the case of a summary, before the scheduled date for the communication and / or presentation of a publication. The medical researcher or doctors will comment on the project within 15 days in the case of a publication and 7 days in the case of a summary, from the date on which the project is received.

However, in the event that the sponsor is in the process of submitting a patent application on the results of the study, the sponsor may delay its publication or communication of the results of the study until the date of registration.

PRO-122 Clinical Trial Protocol: SOPH122-0518 / I Version 1

# 11. Bibliographic references.

- [1] R. Weinreb y P. Khaw, «Primary open-angle glaucoma,» Lancet, vol. 363, pp. 1711-1720, 2004.
- [2] H. Quigley y A. Broman, «The number of people with glaucoma worldwide in 2010 and 2020,» *Br J Ophthalmology*, vol. 90, pp. 262-267, 2006.
- [3] E. Kim y R. Varma, «Glaucoma in Latinos/Hispanics,» *Curr Opin Ophthalmol*, vol. 21, nº 2, pp. 100-105, 2010.
- [4] R. Varma, D. Wang, C. Wu, B. Francis, B. Nguyen, V. Chopra, F. Memarzadeh, M. Torres y S. Azen, «Los Angeles Latino Eye Study Group: Four.year incidence of open-angle glaucoma and ocular hypertension,» *Am J Ophthalmol*, vol. 154, nº 2, pp. 315-325, 2012.

- [5] B. Chauhan, F. Mikelberg, A. Balaszi y C. G. S. Group, «Canadian Glaucoma Study Group: 2. Risk factors for the progression of open-angle glaucoma,» *Arch Ophthalmol*, vol. 126, pp. 1030-1036, 2008.
- [6] Collaborative Normal-Tension Glaucoma Study Group, «Comparison of glaucomatous progression between untreated patients with normal-tension glaucoma and patients with therapeutically reduced intraocular pressures,» *Am J Ophthalmol*, vol. 126, pp. 487-497, 1998.
- [7] M. Kass, D. Heuer y E. Higginbotham, «The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma,» *Arch Ophthalmol*, vol. 120, pp. 701-713, 2002.
- [8] D. Musch, B. Gillespie y L. Nisiol, «CIGTS Study Group. Intraocular pressure control and long-term visual field loss in the Collaborative Initial Glaucoma Treatment Study,» *Ophthalmology*, vol. 118, pp. 1766-1773, 2011.
- [9] A. Heijl, M. Leske y B. Bengtsson, «Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression,» *Arch Ophthalmol*, vol. 120, pp. 1268-1279, 2002.
- [10] P. Bhagat, K. Sodimalla, C. Paul, S. Pandav, G. Raman, R. Ramakrishnan, A. Joshi y A. Raut, «Efficacy and safety of benzalkonium chloride-free fixed dose combination ot latanoprost and timolol in patients with open-angle glaucoma or ocular hypertension,» *Clin Ophthalmol*, vol. 8, pp. 1241-1253, 2014.
- [11] European Glaucoma Society, Terminology and guidelines for glaucoma, Savona, Italia: SvetPrint, 2014.
- [12] S. Sharma, S. Trikha, S. Perera y T. Aung, «Clinical effectiveness of brinzolamide 1%-brimonidine 0.2% fixed combination for primary open-angle glaucoma and ocula hypertension,» *Clin Ophthalmol*, vol. 9, pp. 2201-2207, 2015.
- [13] G. Hollo, F. Topouzis y R. Fechtner, «Fixed-combination intraocular pressure-lowering therapy for glaucoma and ocular hypertension: advantages in clinical practice,» *Expert Opin Pharmacother*, vol. 15, pp. 1737-1747, 2014.
- [14] E. Higginbotham, «Considerations in glaucoma therapy: fixed combinations versus their component medications,» *Clin Ophthalmol*, vol. 4, pp. 1-9, 2010.
- [15] G. Lazcano, A. Hernandez, M. Iriarte y C. Hernandez, «Topical glaucoma therapy cost in Mexico,» *Int Ophthalmol*, vol. 34, pp. 241-249, 2014.
- [16] Y. Goto, N. Ibaraki y K. Miyake, «Human lens epithelial cell damage and stimulation of their secretion of chemical mediators by benzalkonium chloride rather than latanoprost and timolol,» *Arch Ophthalomol*, vol. 121, pp. 835-839, 2003.
- [17] R. Noecker y K. Miller, «Benzalkonium chloride in glaucoma medications,» *Ocul Surf,* vol. 9, nº 3, pp. 159-163, 2011.
- [18] P. Plsella, P. Pouliquen y C. Baudouin, «Prevalence of ocular symptoms and signs with preserved and preservative free glaucoma medication,» *Br J Ophthalmol*, vol. 86, pp. 418-423, 2002.

- [19] J. Cheng, S. Cheng, L. Gao, G. Lu y R. Wei, «Intraocular pressure-loweing effects of commonly used fixed combinations drugs with timolol: a systematic review and meta-analysis,» *PLOS One*, vol. 7, nº 9, pp. e45079-e45090, 2012.
- [20] P. Freeman y M. Kahook, «Preservatives in topical ophtalmic medications: Historical and clinical perspectives,» *Expert Rev Ophthalmol*, vol. 4, nº 1, pp. 59-64, 2009.
- [21] C. Baudouin, P. Pisella, K. Fillacier y e. al., «Ocular surface inflammatory changes induced by topical antiglaucoma drugs: human and animal studies,» *Ophthalmology*, vol. 106, nº 3, pp. 556-563, 1999.
- [22] R. Noecker, L. Herrygers y R. Anwaruddin, «Corneal and conjunctival changes caused by commonly used glaucoma medications,» *Cornea*, vol. 23, pp. 490-496, 2004.
- [23] L. Baiza, J. Álvarez, A. Contreras, J. Medrano, A. De Luca, M. Cortés, M. Garcidueñas, B. Gómez, F. Gil, C. Hartleben, J. Jiménez, M. Moreno, J. Paczka, G. Velasco y M. Vergara, «The efficacy and safety of two fixed combinations: Timolol-dorzolamide-brimonidine versus timolol-dorzolamide. A prospective, randomized, double-masked, multi-center, 6-month clinical trial,» Ann Ophthalmol, vol. 41, pp. 174-178, 2009.
- [24] L. Baiza, J. Llamas y C. Ayala, «Comparison of timolol 0.5% + brimonidine 0.2% + dorzolamide 2% versus timolol 0.5% + brimonidine 0.2% in a Mexican population with primary open-angle glaucoma or ocular hypertension,» *Clin Ophthalmol*, vol. 6, pp. 1051-1055, 2012.
- [25] L. Baiza, J. Alvarez, A. Contreras, J. Medrano, H. Casab, M. Cortés y a. et, «The efficacy and safety of two fixed combinations: timolol-dorzolamide-brimonidine versus timolol-dorzolamide. A prospective, randomized, double-masked, multi-center, 6-month clinical trial,» *Annals of Ophthalmology*, vol. 41, nº 3, pp. 174-178, 2009.
- [26] A. García, J. Paczka, J. Jiménez y C. Hartleben, «Efficacy and tolerability of fixed-combination bimatoprost/timolol versus fixed-combination dorzolamide/brimonidine/timolol in patients with primary open-angle glaucoma or ocular hypertension: a multicenter, prospective, crossover study,» BMC Ophthalmology, pp. 1-12, 2014.
- [27] Laboratorios Sophia, SA de CV, «http://www.medicamentos.com.mx/DocHTM/17147.htm,» Información para prescribir. Producto IMOT OFTENO ( Maleato de timolol 0.5%), [En línea]. Available: http://www.medicamentos.com.mx/DocHTM/17147.htm. [Último acceso: 8 abril 2016].
- [28] Laboratorios Sophia, SA de CV, «http://www.medicamentos.com.mx/DocHTM/20625.htm,» Información para prescribir. Producto Agglad Ofteno (tartrato de brimonidina 0.2%), [En línea]. Available: http://www.medicamentos.com.mx/DocHTM/20625.htm. [Último acceso: 8 abril 2016].
- [29] Laboratorios Sophia, SA de CV, «http://mx.prvademecum.com/producto.php?producto=13288,» Información para prescribir. Producto IOPZOX OFTENO (Dorzolamida 2%), [En línea]. Available: http://mx.prvademecum.com/producto.php?producto=13288. [Último acceso: 8 abril 2016].
- [30] R. Sampaolesi, J. Sampaolesi y J. Zarate, The Glaucomas. Volume II Open Angle Glaucoma and Angle Closure Glaucoma, Buenos Aires, Argentina: Springer, 2014.

- [31] Laboratorios Sophia, SA de CV, «Formulación Krytantek Ofteno Departamento de Investigación y Desarrollo de Laboratorios Sophia S.A. de C.V.,» Gerencia de Desarrollo Farmacéutico, Zapopan, Jalisco, 2007.
- [32] Departamento de Desarrollo Farmacéutico de Laboratorios Sophia S.A. de CV, «Información de Medicamento en Investigación PRO-122,» Fecha de emisión del documento: 14/Mar/16 Gerencia de Desarrollo Farmacéutico, Zapopan, Jalisco, 2016.
- [33] L. Gordis, «General concepts for use of markers in clinical trials,» *Control Clin Trials*, vol. 5, pp. 481-487, 1984.
- [34] M. Mattson y L. Friedman, «Issues in medication adherence assessment in clinical trials of the National Heart, Lung, and Blood Institute,» *Control Clin Trials*, vol. 5, pp. 488-496, 1984.
- [35] S. Norell, «Methods in assessing drug compliance,» *Acta Med Scand*, vol. S 683, pp. 34-50, 1984.
- [36] P. Rudd, R. Byyny, V. Zachary y e. al, «Pill count measures of compliance in a drug trial: variability and suitability,» *Am J Hypertens*, vol. 1, pp. 309-312, 1988.
- [37] K. Farmer, «Methods for measuring and monitoring medication regimen adherence in clinical trials and clinical practice,» *Clin Ther*, vol. 21, pp. 1074-1090, 1999.
- [38] H. Liu, C. Golin, L. Miller y e. al, «A comparison study of multiple measures of adherence to HIV protease inhibitors,» *Ann Intern Med*, vol. 134, pp. 968-977, 2001.
- [39] W. Lam y P. Fresco, «Medication Adherence Measures: An Overview,» *BioMed Research International*, vol. 2015, 2015.
- [40] M. Vitolins, C. Rand, S. Rapp, P. Ribisl y M. Sevick, «Measuring Adherence to Behavioral and Medical Interventions,» *Controll Clin Trial*, vol. 21, pp. 188S-194S, 2000.
- [41] J. Lee, K. Grace, T. Foster, M. Crawley y e. al, «How should we measure medication adherence in clinical trials and practice?,» *Ther and Clin Risk Manag*, vol. 3, nº 4, pp. 685-690, 2007.
- [42] J. Kanski, Oftalmología Clínica, Barcelona: Elsevier, 2009.
- [43] M. Michel, W. Sickenberg y H. Pult, «The effectiveness of questionnaires in the determination of contact lens induced dry eye,» *Ophthal Physiol Opt*, vol. 29, pp. 479-486, 2009.
- [44] N. Efron, «Grading scales for contact lens complications,» *Ophtalmic Physiol Opt,* vol. 18, pp. 182-186, 1998.
- [45] European Group of Graves Orbitopathy, «Eugogo,» ETA, [En línea]. Available: http://www.eugogo.eu/\_downloads/clincial\_evaluation/CHEMOSIS-GO.pdf. [Último acceso: 11 Abril 2016].
- [46] International Dry Eye WorkShop 2007, «Methodologies to diagnose and monitor dy eye disease,» *Ocul Surf*, vol. 5, nº 2, pp. 108-152, 2007.
- [47] A. Haffajee, S. Socransky and J. Lindhe., "Comparison of statistical methods of analysis of data from clinical periodontal trials.," *Journal of Clinical Periodontology*, vol. 10, pp. 247-256, 1983.

- [48] R. Woolson, "Wilcoxon signed-rank test.," Wiley Encuclopedia of Clinical Trials., pp. 1-3, 2008.
- [49] N. Salkind, Encyclopedia of research desing, Thousand Oaks, CA: SAGE Publications Ltd, 2010.
- [50] B. Klingenberg and A. Agresti, "Multivariate extension of McNemar's test.," *Biometrics.*, vol. 62, pp. 921-928, 2006.
- [51] Secretaría de Salud México, «NORMA Oficial Mexicana NOM-220-SSA1-2012, Instalación y operación de la farmacovigilancia.,» *Diario Oficial*, 2013.
- [52] International Conference on Harmanisation of Technical Requirements for Registration of Pharmaceuticals for Human Use, «Clinical Safety Data Management: Definitions and Standards for Expedited Reporting E2A,» *ICH Harmonised Tripartite Guideline*, vol. 4 version, 1994.
- [53] International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use, «General Considerations for Clinical Trials,» *ICH Topic E8*, 1998.
- [54] I. Aramendi, L. Ardao, M. Oyarzun, M. Pérez, I. Olmos y M. Frontini, «Problemas relacionados con medicamentos en pacientes hospitalizados en el Hospital Vilardebó,» *Rev Psiquiatr Urug*, vol. 75, nº 2, pp. 123-133, 2011.
- [55] R. Meyboom, A. Egberts, I. Edwards, Y. Hekster, F. Koning y Gribnau, «Principles of signal detection in pharmacovigilance.,» *Drug Safety*, vol. 16, pp. 355-365, 1997.

# 12. Signature page.

12.1 Signatures of the sponsor's representatives.

| First name: | |
|-----------------------------------|-----------|
| Dr. Leopoldo Martín Baiza Durán | Signature |
| Title: | |
| Medical responsible for the study | Date |
| First name: | |
| QFB. Francisco García Vélez | Signature |
| Title: | |
| Director of the study | Date |

| First name: | |
|--------------------------|-----------|
| Dr. Oscar Olvera Montaño | Signature |
| Title: | |
| Protocol author | Date |

## 12.2 Investigator.

I agree to conduct this clinical study according to the design and guidelines of this protocol, abiding by the provisions of this protocol. I agree to conduct the study in accordance with the accepted standards of Good Clinical Practices. I agree to report all information or data in accordance with what is stated in the protocol, in particular, any adverse event. Also, I agree to handle the clinical supplies, provided by the sponsor, strictly in accordance with this protocol. I understand that the information that identifies me may be used by the sponsor. Because the information contained in this protocol and the Investigator's Manual is confidential, I understand that it is prohibited to share it with any third party, who is not involved in the approval, supervision or conduct of the study. I will make sure to take the necessary precautions to protect information from loss, inadvertent disclosure or access by unauthorized third parties.

| First name: | | |
|-------------|---|-----------|
| | - | Signature |
| Title: | | lly left |
| | | Date |

# 13. Annexes.

# 13.1 Ocular comfort index.

| Identificat | tion file. | | | | | | |
|---|---|---|---|---|---|---|---|
| Study nun | nber <u>SOPH</u> | 122-0518-I | | | Date: | | |
| Initials of | the subjec | t: | | | Subjec | t number | |
| Indications: This questionnaire was designed to qualify the comfort of your eyes. Circle your answer for each question. | | | | | | | |
| Example: | The last we | eek, how oft | en your eye | s were re | ed? | | |
| | Never | | | | <u>Always</u> | | |
| | 0 | 1 2 | 3 | 4 | 5 6 | | |
| There are question. | no correct | or incorrec | t answers. D | o not tak | ke too much ti | me in eacl | n |
| 1 | The last w | eek, how ofte | en your eyes | felt dry? | | | |
| | Never | | | | | | Always |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | When you | r eyes felt dn | y, usually, ho | w intense | was the sensat | tion? | |
| | I have not | | | | | | Severe |
| | felt it | | | | | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 2 | The last w | eek, how ofte | en your eyes | felt sandy | ? | | |
| | Never | | | | | | <u>Always</u> |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | When you | r eyes felt sa | ndy, usually, | how inten | ise was the sen | sation? | |
| | I have not | | | | | | Severe |
| | felt it | _ | _ | | | _ | _ |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 3 | | eek, how ofte | en your eyes | telt throb | bing? | | |
| | Never | | | | | | <u>Always</u> |
| | 0 | 1 | 2 | 3 | . 4 | 5 | 6 |
| | | r eyes felt thi | robbing, usua | ally, how i | ntense was the | sensation? | |
| | I have not | | | | | | Severe |
| | <u>felt it</u><br>0 | 1 | 2 | 2 | 4 | 5 | 6 |
| 4 | | eek, how ofte | _ | falt tirad? | | , | 0 |
| 4 | Never | eek, now one | en your eyes | ieit tireu: | | | Always |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| | | r eves felt tin | _ | _ | e was the sens | _ | 0 |
| | I have not | . cycs leit till | cu, usuany, n | OW HITCHS | e was are sells | acion: | Severe |
| | felt it | | | | | | SEVERE |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

5 The last week, how often your eyes felt sore? Never <u>Always</u> 0 2 3 5 6 When your eyes felt sore, usually, how intense was the sensation? Severe felt it 2 3 5 6 6 The last week, how often your eyes felt itchy? <u>Always</u> 6 When your eyes felt itchy, usually, how intense was the sensation? I have not Severe 1 2 3 4 5 6 0

# 13.2 Efron scale for conjunctival hyperemia.



## 13.3 Oxford Scale.

| PANEL | Grade | Criteria |
|-------|-------|-----------------------------------------------|
| A | 0 | Equal to or less than panel A |
| В | I | Equal to or less than panel B, greater than A |
| С | II | Equal to or less than panel C, greater than B |
| D | III | Equal to or less than panel D, greater than C |
| E | IV | Equal to or less than panel E, greater than D |
| >E | V | Greater than panel E |